## STATISTICAL ANALYSIS PLAN

## A RANDOMIZED PHASE II TRIAL OF GEMCITABINE AND NAB-PACLITAXEL VS. GEMCITABINE, NAB-PACLITAXEL, DURVALUMAB AND TREMELIMUMAB AS 1ST LINE THERAPY IN METASTATIC PANCREATIC ADENOCARCINOMA

#### **Protocol CCTG PA.7**

| Prepared by: | <u>Signature</u> | <u>Date</u> |
|-------------------------------------|-------------------|-------------|
| CCTG/Queen's Statistician | Dongsheng Tu | |
| Reviewed by: | <u>Signature</u> | <u>Date</u> |
| CCTG/Queen's<br>Senior Investigator | Chris O'Callaghan | |

August 9, 2019

#### **ABBREVIATIONS**

AE Adverse Event

ALP Alkaline phosphatase ALT Alanine Aminotransferase

AST Serum Glutamic Oxaloacetic Transaminase

BSA Body Surface Area BUN Blood urea nitrogen

CCTG Canadian Cancer Trials Group

C. I. Confidence Interval

CMH Cochran-Mantel-Haenszel

CR Complete Response CRF Case Report Form

CTCAE Common Terminology Criteria for Adverse Events
CTLA-4 Cytotoxic T-lymphocyte-associated protein 4
DSMC Data and Safety Monitoring Committee
ECOG Eastern Cooperative Cancer Group

ECG Electrocardiography

EORTC European Organization for Research and Treatment of Cancer

G+N Gemcitabine and nab-paclitaxel

G+N+D+T Gemcitabine and nab-paclitaxel with durvalumab and tremelimumab

iCPD Immune confirmed progression disease

iCR Immune complete response

IN Inevaluable

INR International Normalized Ratio (for Prothrombin Time)

iPR Immune partial response

irAE Immune Related Adverse Event

iRECIST Immune Response Evaluation Criteria in Solid Tumors

iSD Immune stable disease

iUPD Immune unconfirmed progression disease

LDH Serum Lactate Dehydrogenase LKA Last day the patient is Known Alive

LLN Lower Limit of Normal MPV Major Protocol Violation

NA Not Assessed NC Not Computed

ORR Objective Response Rate

OS Overall Survival PD Progression Disease

PD1 Programmed cell death protein 1 PD-L1 Programmed cell death ligand 1

PFS Progression-free survival

PR Partial Response
PT Prothrombin Time

PTT Partial Thromboplastin Time QLQ Quality of Life Questionnaire

QOL Quality of Life

RBC Red Blood Cell Count

Response Evaluation Criteria in Solid Tumors Statistical Analysis System Stable Disease RECIST

SAS

SD STD Standard Deviation WBC White Blood Cell Count

## TABLE OF CONTENTS

| 1. | В | ackground and Rationale | 7 |
|---|---|---|---|
| 2. | Si | tudy Description | 7 |
| 2 | | Study Design | |
| 2 | | Treatment Allocation | |
| <i>3</i> . | | bjectives | |
| | | Primary | |
| | | Secondary | |
| <i>4</i> . | | ndpoints | |
| 4 | .1 | Primary Efficacy | 9 |
| 4 | .2 | Secondary Efficacy | 9 |
| 4 | .3 | Safety | 9 |
| <i>5</i> . | | ample Size and Power | |
| 6. | | ata Set Descriptions | |
| 7. | | | |
| | | fatistical Analysis | |
| | | General Methods | |
| 7 | .2 | Data Conventions | 11 |
| 7 | | Study Conduct | 11 |
| | 7.3.1 | 1 | $\frac{11}{11}$ |
| | 7.3.2<br>7.3.3 | | $\frac{11}{11}$ |
| 7 | .4 | | |
| , | 7.4.1 | | $-\frac{12}{12}$ |
| | 7.4.2 | | $\frac{12}{12}$ |
| | 7.4.3 | | |
| | 7.4.4 | | $-\frac{12}{12}$ |
| | 7.4.5 | | 12 |
| | 7.4.6 | Baseline Exams | 13 |
| | 7.4.7 | | 13 |
| 7 | .5 | Extent of Exposure | 13 |
| | 7.5.1 | Study Therapy | 13 |
| | 7.5.2 | Dose Reduction, Omission, Discontinuation, or IV Rate Decrease or Infusion | |
| | | ruption | 14 |
| | 7.5.3 | Cumulative Dose, Dose Intensity and Relative Dose Intensity | 14 |
| | 7.5.4 | Off Study Therapy | 14 |
| 7 | .6 | Efficacy | 15 |
| | 7.6.1 | Overall survival | 15 |
| | 7.6.2 | Overall Survival by Subsets | 16 |
| | 7.6.3 | Progression-free Survival | 16 |
| | 7.6.4 | Progression-free survival by Subsets | 17 |
| | 7.6.5 | Treatment Objective Response | 17 |
| | 7.6.6 | Treatment Objective Response by Subsets | 17 |

| 7.6.7 | Duration of Objective Response | 18 |
|---|---|---|
| 7.6.8 | Treatment Immune Response (iRECIST) | 18 |
| 77 0 | afata. | 10 |
| | afety | |
| 7.7.1<br>7.7.2 | Adverse Events | 10 |
| | 2.1 Hematology | |
| 7.7.2 | 2.3 Thyroid Function Tests | $\frac{20}{20}$ |
| 7.7.3 | 2.3 Coagulation | $\frac{20}{20}$ |
| 7.7.3 | Other Safety | $\frac{20}{20}$ |
| | 3.1 ECG | $\frac{20}{20}$ |
| 7.7.4 | Deaths on Study/Adverse Events Leading to Discontinuations of Protocol T | |
| /./. <del>4</del> | Deaths of Study/Adverse Events Leading to Discontinuations of Flotocol 1 | reatment 20 |
| 7.8 C | Concomitant Medications, Other Anti-Cancer Treatments, and Majo | r Medical |
| Problen | 18 | 20 |
| 7.9 Q | | 21 |
| 7.9 Q | Quality of Life | |
| 7.9.1 | EORTC QLQ-C30 | 21 |
| 7.9.2 | Data Sets | 22 |
| | Compliance Primary Analysis of COL | |
| 7.9.4 | Primary Analyses of QOL | 22 |
| 7.9.5 | Baseline and Change Score Analysis | 22 |
| 7.9.6 | QOL Response Analysis | 23 |
| 8. Api | pendices | 24 |
| | dix 1: Tables and Figure | |
| | atient Disposition | |
| | ollow-up of Patients | |
| | ccrual by Center | |
| | ccrual by Stratification Factor at Randomization | |
| | ligibility and Reasons for Ineligibility and Major Protocol Violations | |
| Table 6: Tr | reatment as Randomized Versus as Treated | 26 |
| Table 7: Pi | retreatment Characteristics at Baseline | 27 |
| | rior Surgery | |
| Table 9: Pi | rior Radiotherapy | 28 |
| | Prior Systemic Therapy | |
| | Extent of Disease (Target Lesions) | |
| | Extent of Disease (Non-Target Lesions) | |
| | Baseline Signs and Symptoms | |
| | Baseline Hematology | |
| | Baseline Chemistry | |
| | Baseline Thyroid Function Tests | |
| | Baseline Coagulation Tests | |
| | Baseline ECG | |
| | Baseline Urinalysis | |
| | Concomitant Medications at Baseline | |
| | Major Medical Problems at Baseline | |
| | Number of Patients by Cycle | |
| | Number of Cycles of Protocol Therapy per Patient | |
| | Total Treatment Duration | |
| | Dose Reduction, Omission or Delay and Infusion Interruption | |
| 1able 26: ( | Cumulative Dose | 40 |

| Table 27: | Dose Intensity | 40 |
|---|---|---|
| | Relative Dose Intensity | |
| | Off Treatment Summary | |
| | All Deaths | |
| Table 31: | Log Rank and Cox Regression Model for Overall Survival | 43 |
| | Survival by Subsets | |
| | Progression Summary | |
| Table 34: | Log Rank and Cox Regression Model for Progression Free Survival (PFS) | 45 |
| Table 35: | Progression Free Survival (PFS) by Subsets | 46 |
| | Treatment Objective Response | |
| Table 37: | Cochran Mantel Haenszel and Logistic Regression Model for Objective Response | 48 |
| Table 38: | Objective Response According to Pretreatment Characteristics | 49 |
| | Duration of Objective Response | |
| | Immune Response (iRECIST) | |
| | Cochran Mantel Haenszel and Logistic Regression Model for Immune Response | |
| | Immune Response According to Pretreatment Characteristics | |
| | Duration of Immune Response | |
| | Acute (On Treatment) Adverse Events | |
| | Severe Acute (On Treatment) Adverse Events | |
| | Drug Related Acute (on Treatment) Adverse Events | |
| | Immune-related Acute (On Treatment) Adverse Events | |
| Table 48: | Severe Acute (On Treatment) Immune-related Adverse Events | 57 |
| | Delayed (During Follow-up) Adverse Events | |
| | Hematology During Protocol Treatment: Worst Grade per Patient | |
| | Hematology During Follow-up: Worst Grade per Patient | |
| | Serum Chemistry during Protocol Treatment: Worst Grade per Patient | |
| | Serum Chemistry During Follow-up: Worst Grade per Patient | |
| | Thyroid Function Tests: Worst During Protocol Treatment | |
| Table 55: | Thyroid Function Tests: Worst during Follow-up | 68 |
| Table 56: | Coagulation Tests: Worst During Protocol Treatment | 69 |
| | Coagulation Tests: Worst During Follow-up | |
| Table 58: | ECG Results During Protocol Treatment | 70 |
| Table 59 | : Urinalysis During Protocol Treatment | 70 |
| | Deaths During or within 4 weeks of Last Protocol Treatment | |
| Table 61: | Adverse Event leading to Discontinuation of protocol Treatment <sup>(a)</sup> | 71 |
| Table 62: | Concomitant Medications | 71 |
| Table 63: | Anti-Cancer Treatment | 72 |
| Table 64: | Major Medical Problems | 72 |
| Table 65: | Compliance Rate with QoL Assessment by Treatment Arm | 73 |
| Table 66: | Proportion of Patients with Deterioration, Improvement or Stable QoL | 73 |
| Table 67: | Time to Deterioration in QoL Primary Endpoints | 74 |
| Table 68: | QoL: Summary Baseline Scores | 74 |
| Table 69: | Summary QOL Change Scores from Baseline for Scale/Domain/Item at Each Time Pe | riod* |
| | | 75 |
| Table 70: | Results for QOL Response Analyses | 76 |
| | <u>Figures</u> | |
| Figure 1. | Accrual by Calendar Time | 25 |
| Figure 2: | Kaplan-Meier Curves for Overall Survival | 42 |
| | Kaplan-Meier Curves for Progression Free Survival | |

## 1. Background and Rationale

The purpose of this document is to describe the analysis of PA.7 for the writing of a Canadian Cancer Trials Group (CCTG) study report on this study. The data are collected and cleaned by CCTG. All analyses will be performed by a senior biostatistician in CCTG and a final statistical analysis report will be prepared. A copy of this report will be sent to the study chair for the writing of the manuscript and to AstraZeneca.

#### **Rationale of the Study:**

Programmed cell death ligand 1 (PD-L1), the ligand for programmed cell death protein 1 (PD1), is part of a complex system of receptors and ligands that are involved in controlling T-cell activation, which acts at multiple sites in the body to help regulate normal immune responses and is utilized by tumours to help evade detection and elimination by the host immune system. In a number of cancers including pancreatic cancer, overexpression of PD-L1 is associated with reduced survival and unfavourable prognosis. Clinically, blockade of the PD-1 inhibitory checkpoint pathway by inhibiting PD-L1/PD-1 engagement has been shown to induce tumour regression across many cancer types, including melanoma and renal cell, colon and lung cancers. CTLA-4 is another co-inhibitory receptor expressed on activated T cells and regulates early stage T cell activation, reducing the amplitude of T-cell activation. Targeting both PD-1 and CTLA-4 pathways may have additive or synergistic activity because the mechanisms of action of CTLA-4 and PD-1 are non-redundant. This study was designed to evaluate whether combining PD-1/PD-L1 and CTLA-4 inhibition with durvalumab and tremelimumab will lead additional benefits to standard 1st line chemotherapy with gemcitabine/nab-paclitaxel in metastatic pancreatic cancer.

#### **Research Hypothesis:**

The primary hypothesis in this study is that durvalumab and tremelimumab combined with standard 1st line chemotherapy with gemcitabine/nab-paclitaxel (Arm G+N+D+T) will have a greater clinical efficacy compared to standard 1st line chemotherapy with gemcitabine/nab-paclitaxel (Arm G+N) in patients with metastatic pancreatic cancer as measured by overall survival.

#### **Schedule of Analyses:**

Only one analysis will be performed, when 150 events (deaths) have been observed.

## 2. Study Description

## 2.1 Study Design

PA.7 is an open-label, randomized, non-blinded, phase II clinical study of durvalumab+tremelimumab in combination with gemcitabine and nab-paclitaxel (Arm G+N+D+T) versus gemcitabine and nab-paclitaxel (Arm G+N) in patients with newly diagnosed, untreated, metastatic pancreatic adenocarcinoma. Prior to the randomized component, 10 patients would first be accrued to ensure safety and tolerability of the combination. After the safety profile of these patients was assessed, 180 patients would be randomized in a 2:1 ratio to Arm G+N+D+T or G+N after stratification by ECOG

performance status (0 vs. 1) and receipt of prior adjuvant therapy (yes versus no). Overall survival (OS) was the primary endpoint of this study. The study was conducted by the Canadian Cancer Trials Group (CCTG), with the support of AstraZeneca. CCTG Case Report Forms (CRFs) are used and the database are maintained by CCTG.

This study opened to accrue patients on August 22, 2016. Accrual to safety run-in component of the study was completed on January 23, 2017 with a total of 11 patients enrolled. The first analysis of the run-in patients was performed in March 2017 when all of the patients completed at least one cycle of treatment and, after the review of the results, accrual to randomized Phase II component was opened on April 10, 2017. With permission from the DSMC, an analysis was performed in the middle of January 2018 on a database locked on January 12, 2018 to generate tables and figures for the internal planning of AstraZeneca. The results of this analysis were also presented to DSMC at beginning of February 2018 with a proposal to transition the trial to phase III by CCTG. After reviewing the results, DSMC Chair recommended to continue the phase II trial as currently designed and place the transition "on hold". This recommendation was affirmed by DSMC after reviewing an updated analysis at their 2018 Annual Spring Meeting in April 2018. The accrual of the trial was closed on July 28, 2018 after its accrual goal of 180 patients has been achieved. At its Fall Teleconference in November 2018, the DSMC reviewed a request by the trial team to support an unplanned interim analysis based on the endpoint of overall survival when 100 deaths had occurred for the purpose of informing a potential phase III study design. After reviewing the response to questions raised during the review, this request was approved by the DSMC on March 18, 2019. The analysis was performed at end of April 2019 on a database locked on April 12, 2019 after all deaths observed before April 8, 2019 were reviewed. DSMC recommended the trial continue on to its final analysis as planned after reviewing the results of this analysis at its meeting on May 3, 2019. This analysis plan describes the analyses performed for the final analysis planned when 180 events are observed.

The CCTG Data Safety Monitoring Committee has been reviewing safety data every six months (usually at the time of the bi-annual CCTG Spring and Fall meetings) and as otherwise required. These analyses have been prepared by a CCTG/Queen's Senior Biostatistician.

#### 2.2 Treatment Allocation

The study is planned to randomize 180 subjects using a 2:1 allocation to durvalumab and tremelimumab in combination with gemcitabine and nab-paclitaxel (G+N+D+T Arm) and gemcitabine and nab-paclitaxel alone (G+N Arm). The randomization was dynamically balanced by ECOG performance status (0 vs. 1) and receipt of prior adjuvant therapy (yes versus no) using the method of minimization. A centralized system was used to randomize all patients in this study.

### 3. Objectives

### 3.1 Primary

The primary objective of this study is to compare overall survival of patients with metastatic pancreatic cancer treated with durvalumab and tremelimumab combined with gemcitabine and nab-paclitaxel to the overall survival of patients treated with gemcitabine and nab-paclitaxel alone.

#### 3.2 Secondary

Secondary objectives are to:

- Compare progression-free survival (PFS) between the two treatment arms.
- Compare objective response rates (ORR) between the two treatment arms.
- Assess the toxicity and safety profile of the combination of durvalumab and tremelimumab with gemcitabine and nab-paclitaxel.

### 4. Endpoints

#### 4.1 Primary Efficacy

The primary efficacy endpoint is overall survival.

#### 4.2 Secondary Efficacy

The secondary efficacy endpoints are progression-free survival and objective response rate.

#### 4.3 Safety

The safety endpoints are serious and non-serious adverse events (clinical and laboratory), laboratory parameters, dosing data (including dose interruptions, total delivered dose and dose modifications) and reasons off treatment.

## 5. Sample Size and Power

The primary objective of this study is to assess the additional effect of durvalumab and tremelimumab to gemcitabine and nab-paclitaxel by comparing overall survival (OS) between G+N+D+T and G+N Arms among all randomized patients. It was calculated that with a 2-sided alpha of 10%, a total of 180 patients with 150 events (deaths) would be required to provide 80% power to detect a 4.6 month difference in median survival (a hazard ratio of 0.65) between the two treatment arms assuming a median survival of 8.5 months for the gemcitabine and nab-paclitaxel alone arm. The final analysis will be conducted after at least 150 events have been recorded. It is estimated that 180 patients accrued over 18 months and followed for 17 months will be required to reach the necessary number of events.

## 6. Data Set Descriptions

Three types of analysis samples will be used:

#### All Randomized Patients:

All patients who have been randomized in the study with the treatment arm being as randomized.

#### Response-Evaluable Patients:

All patients who have received at least one cycle of therapy and have their disease reevaluated will be considered evaluable for response (exceptions will be those who exhibit objective disease progression prior to the end of cycle 1 who will also be considered evaluable).

#### All Treated Patients:

All patients who received at least one dose of protocol treatment. Patients randomized to G+N Arm who have received at least one dose of durvalumab and tremelimumab on study (from Cancer Treatment Section of Treatment Report) will be grouped with patients randomized to G+N+D+T in the analyses of safety.

## 7. Statistical Analysis

#### 7.1 General Methods

All comparisons between treatment arms will be carried out using a two-sided test at an alpha level of 10% unless otherwise specified.

When appropriate, discrete variables are summarized with the number and proportion of subjects falling into each category, and compared using Fisher's exact test. Continuous and ordinal categorical variables are summarized using the mean, median, standard error, minimum and maximum values and when appropriate, compared using the Wilcoxon test. All confidence intervals are computed based on normal approximations except those for rates, which will be computed based on the exact method

Time to event variables are summarized using Kaplan-Meier plots. Primary comparisons of the treatment groups are made using the stratified log-rank test. Primary estimates of the treatment differences are obtained with the hazard ratios and 90% confidence intervals from stratified Cox regression models using treatment arm as the single factor.

Percentages given in the summary tables will be rounded and may therefore not always add up to exactly 100%. Listings, tabulations, and statistical analyses will be carried out using the SAS (Statistical Analysis System, SAS Institute, North Carolina, USA) software.

Unless otherwise specified, date of randomization and stratification factors will be taken from the Centralized Randomization File.

Baseline evaluations will be those collected on Eligibility Checklist and Baseline Report and closest to, but no later than, the first day of study medication for treated subjects and closest to, but no later than, the date of randomization, for subjects who were randomized but who never received treatment.

Laboratory results, adverse events, and other symptoms are coded and graded using the Common Terminology Criteria for Adverse Events (CTCAE v4.0).

#### 7.2 Data Conventions

When converting a number of days to other units, the following conversion factors will be used:

```
1 year = 365.25 days
1 month = 30.4375 days
```

When either day or month of a date is missing, the missing day and/or month will be imputed by the midpoint within the smallest known interval. For example, if the day of the month is missing for any date used in a calculation, the 15th of the month will be used to replace the missing day. If the month and day of the year are missing for any date used in a calculation, the first of July of the year will be used to replace the missing date.

#### 7.3 Study Conduct

All randomized patients are included in the analyses of study conduct. Information will be tabulated by randomized treatment (unless otherwise indicated) and pooled treatments.

#### 7.3.1 Patient Disposition

- Number of patients randomized, treated (on study, off study), never treated (Table
   1)
- Number of alive patients (Table 2)
- Median (estimated by Kaplan-Meier method) and range (minimum and maximum)
  (Table 2) of the follow-up time (months) defined as time from the day of
  randomization (as recorded in centralized randomization file) to the last day the
  patient is known alive (LKA) as the last recorded date known alive or censored at
  the time of death and calculated as

[(date of death or LKA – date of randomization) + 1)]/30.4375.

#### 7.3.2 Accrual Patterns

- Number of patients randomized by center (**Table 3**)
- Number of patients by stratification factors at randomization (**Table 4**)
- Accrual of patients by calendar time pooled across two treatment arms (Figure 1)

#### 7.3.3 Eligibility Violations/Protocol Deviations

Eligibility violations of inclusion or exclusion criteria are centrally reviewed by CCTG; a field (y/n) for eligibility status and reason for ineligibility is entered in the database. A major protocol violation (MPV) is defined as a deviation from the protocol, initiated by the centre or the investigator, serious enough to mean that the patient's data

contributes little, if any, information on the efficacy or toxicity of the regimen under study. MPVs are coded by CCTG based on its standard codes.

- Number of patients eligible, not eligible (Table 5)
- Reasons for ineligibility (**Table 5**)
- Major protocol violations: % for each type of violations (**Table 5**).

Deviations from randomization will be summarized as follows:

• Treatment as randomized versus as treated (**Table 6**)

#### 7.4 Study Population

All randomized patients are included in the study population analyses. Information will be tabulated by randomized treatment (unless otherwise indicated) and pooled treatments.

#### 7.4.1 Patient Pretreatment Characteristics

- Gender (Table 7)
- Race (Table 7)
- Age: median, minimum, maximum values; number <65, ≥65 (**Table 7**)
- ECOG Performance Status: 0, 1 (**Table 7**)
- BSA: median, minimum, maximum values (**Table 7**)
- Months from initial diagnosis of pancreatic cancer to randomization: median, minimum, maximum values (Table 7)
- Metastatic disease at initial diagnosis: Yes, No (Table 7)
- Months from diagnosis of metastatic disease following completion of prior surgical/adjuvant therapy: median, minimum, maximum values (**Table 7**)

#### 7.4.2 Prior Surgery

- Number of patients with prior surgery for colorectal cancer (**Table 8**)
- Procedure/site of prior surgery (Table 8)

#### 7.4.3 Prior Radiotherapy

- Number of patients with prior radiotherapy for pancreatic cancer (Table 9)
- Prior radiotherapy by site (**Table 9**)

#### 7.4.4 Prior Systemic Therapy

- Number of subjects with prior systemic therapy and type of prior systemic therapy (adjuvant, metastatic, neo-adjuvant) (Table 10)
- Number of patients with specific drug/agent (Table 10)

#### 7.4.5 Extent of Disease

- Number of patients with target lesions, number of target lesions, largest measure, site of target lesions (**Table 11**)
- Number of patients with non-target lesions, number of non-target lesions, site of non-target lesions (Table 12)

#### 7.4.6 Baseline Exams

- Baseline signs and symptoms (**Table 13**)
- Baseline hematology: WBC, neutrophils, platelets, hemoglobin, RBC, lymphocytes, monocytes, eosinophils, basophils (**Table 14**)
- Baseline serum chemistry: Total bilirubin, AST, ALT, LDH, creatinine clearance, serum creatinine, chloride, sodium, albumin, potassium, calcium, magnesium, ALP, glucose, amylase, lipase, Urea, BUN (**Table 15**)
- Baseline Thyroid Function Tests (Table 16)
- Baseline Coagulation Tests (**Table 17**)
- Baseline ECG (Table 18)
- Baseline urinalysis (Table 19)

#### 7.4.7 Concomitant Medications and Major Medical Problems at Baseline

- Number of patients with concomitant medication within 14 days prior to the date of randomization (**Table 20**)
- Number of patients with past or current major medical problems ongoing at baseline (Table 21)

#### 7.5 Extent of Exposure

Patients included are those who received at least one dose of protocol treatment as defined in Section 6.

#### 7.5.1 Study Therapy

During a 4 week cycle of protocol treatment, the patients on both arms would receive infusion of gemcitabine (1000 mg/m<sup>2</sup>) and nab-paclitaxel (125 mg/m<sup>2</sup>) on days 1, 8 and 15. Patients on G+N+D+T arm would receive in addition infusion of durvalumab (1500 mg) on day 1, and tremelimumab (75 mg) on day 1 of cycles 1, 2, 3 and 4 only.

Duration of gemcitabine or nab-paclitaxel (in weeks) during the study is defined as follows:

[last date of infusion of gemcitabine or nab-paclitaxel – first date of infusion of gemcitabine or nab-paclitaxel + 14]/7,

where the first and last date of infusion is taken from Gemcitabine Administration or Nab-paclitaxel Administration Section of Treatment Report.

Duration of durvalumab or tremelimumab (in weeks) during the study is defined as follows:

[last date of infusion of durvalumab or tremelimumab – first date of infusion of durvalumab or tremelimumab + 28]/7,

where the first and last date of infusion is taken from Durvalumab Administration or Tremelimumab Administration Section of Treatment Report).

The following variable will be summarized using the data set of all treated patients:

- Number of patients by cycle of therapy (Table 22)
- Total number of cycles of treatment per patient (Table 23)
- Total treatment duration per patient for each drug (Table 24)

# 7.5.2 Dose Reduction, Omission, Discontinuation, or IV Rate Decrease or Infusion Interruption

The administration of protocol treatment in a cycle may be modified (delayed, omitted, reduced, and infusion interrupted) because of toxicity or other reasons. For each drug, the following variables will be summarized using the data set of all treated patients:

- Number of patients with at least one cycle reduced, omitted, delayed, or infusion interrupted (Table 25)
- Reason for these dose modifications (Table 25)

#### 7.5.3 Cumulative Dose, Dose Intensity and Relative Dose Intensity

The cumulative dose (mg) per patient for durvalumab and tremelimumab is the total dose (mg) that the patient received. The cumulative dose (mg/m²) per patient for gemcitabine and nab-paclitaxel is defined as the sum over all cycles of the total actual dose received divided by the BSA in a given cycle (**Table 26**).

The actual dose intensity of a drug (mg/week) per patient is defined as:

Actual Dose Intensity = 
$$\frac{\text{Cumulative dose } (\frac{\text{mg}}{m^2} \text{ or mg})}{\text{Duration of treatment}}.$$

where duration of treatment is defined in 7.5.1 (**Table 27**).

The relative dose intensity per patient for each drug is defined as the dose intensity (mg/m²/week or mg/week) divided by the planned weekly dose as assigned in the protocol, which is 375 mg/week for durvalumab, 18.75 mg/week for tremelimumab, 750 mg/m²/week for gemcitabine, and 93.75 mg/m²/week for nab-paclitaxel.

The patient relative dose intensities will be grouped according to the following categories: <60%,  $\ge 60\%$ ,  $\ge 80\%$ ,  $\ge 80\%$ ,  $\ge 90\%$ , (**Table 28**).

#### 7.5.4 Off Study Therapy

The reason for off of each study therapy will be taken from End of Treatment Section of End of Treatment Report.

The following information will be summarized for each of protocol treatment (**Table 29**):

- Number of patients off study treatment
- Reason off protocol therapy

#### 7.6 Efficacy

#### 7.6.1 Overall survival

For all randomized patients, survival is calculated from the day of randomization (as recorded in Centralized Randomization File) to death (Date/Cause of Death Section of Death Report). For alive patients, survival is censored at the last day the patient is known alive (LKA) as the last recorded date known alive (last date of infusion of gemcitabine, nab-paclitaxel, durvalumab or tremelimumab in Treatment Report, Date of Attendance/Last Contact on 4-Week Post Treatment Report, Follow-up Report, Short Follow Up Report, and Minimal Follow-up Report). Survival time (in months) is defined as

[(date of death or LKA – date of randomization) + 1)]/30.4375.

A frequency table for the number of patients who died and cause of death in each treatment arm will be provided (**Table 30**). Kaplan-Meier curve for proportions of survival in each treatment arm will be displayed (**Figure 2**).

The comparison of overall survival between the two treatment arms is the primary objective of this study. The primary analysis will be the log-rank test (**Table 31**) stratified by the factors coded as:

**Stratification Factors (at randomization)** 

Performance status 1 = ECOG 0 0 = ECOG 1Prior adjuvant chemotherapy 1 = Yes 0 = No

The hazard ratio of durvalumab and tremelimumab combined with gemcitabine and nab-paclitaxel (G+N+D+T Arm) over gemcitabine and nab-paclitaxel alone (G+N Arm) and two-sided 90% CI will be calculated (**Table 31**) based on the Cox regression model stratified by above stratification factors, and with treatment arm coded as G+N+D+T Arm=1 and G+N Arm=0. The 90% confidence intervals for the median survival will be computed using the method of Brookmeyer and Crowley [2].

In order to assess the influence of the potential prognostic factors shown and coded below on the comparison of survival between treatment arms, a stratified Cox regression model will be used with all variables (treatment arm and prognostic factors) included to estimate hazard ratios and 90% confidence intervals (**Table 31**).

#### Prognostic factors (at baseline)

| Gender | 0 = Female | 1 = Male |
|-----------------------|--------------|------------|
| Age | $0 = \ge 65$ | 1 = < 65 |
| Number of organ sites | 0 = >2 | $1=\leq 2$ |

No interactions will be considered in the model.

#### 7.6.2 Overall Survival by Subsets

For each level of the following baseline variables, a Kaplan-Meier plot of survival by treatment arm will be produced as well as medians with 90% C.I. and the hazard ratio (unstratified) with 90% CI of durvalumab or tremelimumab combined with gemcitabine and nab-paclitaxel (G+N+D+T Arm) over gemcitabine and nab-paclitaxel alone (G+N Arm) (**Table 32**):

• Gender: male, female

• Age:  $<65, \ge 65$ 

• Race: white, black, other

• Performance status at baseline: ECOG 0, 1

• Number of organ sites involved at baseline:  $\leq 2$  versus  $\geq 2$ 

#### 7.6.3 Progression-free Survival

Progression-free survival (PFS) will be calculated for all patients from the day of randomization until the first observation of disease progression (date of objective relapse or progression of Relapse/Progression Report) or death due to any cause (recorded in Date/Cause of Death Section of Death Report) as the (difference+1).

If a patient has not progressed or died, PFS will be censored on the date of last disease assessment defined as the earliest test date of target lesion or non-target lesions (if patient has no target lesions), whichever is latest.

A frequency table will be provided describing progression and censoring as follows (Table 33):

- Number of patients who progress (documented progression, death without documented progression)
- Number of patients censored (alive and not progressed)

Analyses for PFS will be similar to that for overall survival as previously described. A Kaplan-Meier curve for PFS in each treatment arm will be displayed (**Figure 3**). In the primary analysis, median PFS for the two treatments will be compared using the stratified log-rank test (**Table 34**). A stratified Cox regression model will estimate the durvalumab and tremelimumab combined with gemcitabine and nab-paclitaxel (G+N+D+T Arm) over gemcitabine and nab-paclitaxel alone (G+N Arm) PFS hazard ratio and 90% C. I. (**Table 34**). In addition, a stratified Cox regression model adjusted for covariates will be applied to verify the impact of the prognostic factors on the treatment effect (**Table 34**).

Coding for treatment arm, stratification variables and prognostic factors is identical to that presented in **Section 7.6.1**.

Some patients received other anti-cancer therapy before progression or death. Sensitivity analyses will be performed by censoring those who have received anti-cancer therapy prior to documentation of disease relapse/progression or death on the

earliest date cancer treatment began or treating them as having PFS events at the earliest date when the treatment began.

#### 7.6.4 Progression-free survival by Subsets

Subset analyses performed for overall survival will also be performed for PFS (**Table 35**).

#### 7.6.5 Treatment Objective Response

All patients will have their best objective response on study classified every 8 weeks until disease progression, using the RECIST (Response Evaluation Criteria in Solid Tumors) criteria 1.1. The best response to protocol treatment is collected in "Best Overall Response" section of END OF TREATMENT REPPORT. For patients who are still on protocol treatment and followed for response at final clinical cut-off, their best objective response is defined as the "best verified" objective response they have achieved up to the time of clinical cut-off determined by CCTG Senior Investigator based on data on "Response Assessment" section of TREATMENT REPORT.

Best objective response to protocol treatment will be summarized for all randomized patients (**Table 36**).

The primary analysis of objective response will be the comparison of the objective response rate (CR+PR) between treatment arms among all the randomized patients using the Cochran-Mantel-Haenszel (CMH) statistic adjusted for stratification factor for all randomized patients (**Table 37**) as defined in Section 6.

In addition, a stratified logistic regression model adjusted for covariates will be applied to verify the impact of the prognostic factors on the treatment effect (**Table 37**). For all stratified logistic regression models, estimates of the odds ratio(s) and 90% confidence interval(s) will be given.

Stratified logistic regression odds ratios will be estimated using PROC PHREG in SAS [5]. A dummy time variable will be created, where all responders will be classified as events with an arbitrary time =  $t_0$ , and non-responders as censored with time  $t_1$ , where  $t_1 > t_0$ . The DISCRETE option will be used for tied observations.

Coding for treatment, stratification variable and prognostic factors is identical to that presented in Section 7.4.1.

#### 7.6.6 Treatment Objective Response by Subsets

For all randomized patients, the objective response rate will be presented for each treatment arm in the subgroups defined by the categorical variables listed below (**Table 38**). No formal comparisons are planned:

- gender (male, female)
- age (<65 years,  $\ge65$  years)
- race (white, black, other)

- performance status at baseline (ECOG 0, ECOG 1)
- Number of organ sites involved at baseline ( $\leq 2 \text{ versus} > 2$ ).

#### 7.6.7 Duration of Objective Response

For patients whose best objective responses are classified as CR or PR at any reporting period during the study, the duration of objective response is calculated as the time from CR or PR is documented (whichever is the first) until first observation of objective disease relapse or progression or death due to any cause. If a patient has not relapsed/progressed or died, duration of response will be censored on the date of last disease assessment defined as the earliest test date of target lesion or non-target lesions (if patient has no target lesions), whichever is latest.

All randomized patients with CR or PR are included in this analysis. The median duration of objective response and associated 95% confidence intervals will be computed and compared by the stratified log-rank test adjusting for stratification factors at randomization (Table 39).

#### 7.6.8 Treatment Immune Response (iRECIST)

All patients will also have their response classified every 8 weeks using the modified iRECIST guidelines. The best immune response (iRECIST) to protocol treatment is collected in "Best Objective Response i-RECIST" section of END OF TREATMENT REPPORT. For patients who are still on protocol treatment and followed for response at final clinical cut-off, their best immune response is defined as the "best verified" response they have achieved up to the time of clinical cut-off determined by CCTG Senior Investigator based on data on "Investigator Assessment-i-RECIST" section of TREATMENT REPORT.

All analyses performed for objective response as listed above will be performed similarly for immune response (**Table 40** to **Table 43**).

#### 7.7 Safety

The safety analyses will based on the All Treated population defined in Section 6. Adverse events and laboratories are graded and categorized using the CTCAE v4.0 criteria except where CTCAE grades are not available.

#### 7.7.1 Adverse Events

Adverse events will be recorded on the CCTG toxicity/adverse event-intercurrent illness case report form. Events reported on Treatment Report or 4-Week Post-Treatment Follow-Up Report will be defined as acute (on treatment) adverse events; Events reported on Follow-up Report or Short Follow-up Report will be defined as delayed adverse events.

Drug related adverse events are those events with a relation to protocol therapy of 3=possible, 4=probable or 5=definite.

Severe adverse events are those events reported with a CTCAE Grade of 3 or higher.

Comparisons between treatment arms on acute adverse events (any vs. other, severe vs. other) will be carried out using a two sided Fisher's exact test at an alpha level of two-sided 10%.

The following variables are summarized. Tabulations of overall adverse events will be presented by treatment group.

- Acute Adverse events: worst CTCAE grade per patient (Table 44)
- Severe acute adverse events: worst CTCAE grade per patient (Table 45)
- Drug related acute adverse events: worst CTCAE grade per patient (Table 46)
- Immune-related acute adverse event: worst CTCAE grade per patient (**Table 47**)
- Severe immune-related acute adverse event: worst CTCAE grade per patient (Table 48)
- Delayed adverse events: worst CTCAE grade per patient (**Table 49**)

#### 7.7.2 Laboratory Evaluations

Laboratory evaluations reported on Treatment Report or 4-Week Post-Treatment Follow-Up Report will be included in the calculation for acute (on treatment) laboratory adverse events. All laboratory evaluations reported on Follow-up Report or Short Follow-up Reports will be included in the calculation for delayed (during follow-up) laboratory adverse events. Laboratory results will be classified according to CTCAE version 4.0. Laboratory tests that are not covered by the CTCAE grading system will be summarized according to the following categories: normal and above the upper normal limits.

#### 7.7.2.1 Hematology

- Hemoglobin, platelets, WBC, neutrophils, RBC, lymphocytes, monocytes, eosinophils, basophils on treatment: worst CTC grade per patient (Table 50)
- Hemoglobin, platelets, WBC, neutrophils, RBC, lymphocytes, monocytes, eosinophils, basophils during follow-up: worst CTC grade per patient (Table 51)

#### 7.7.2.2 Serum Chemistry

- Total bilirubin, AST, ALT, LDH, creatinine clearance, serum creatinine, chloride, sodium, albumin, potassium, calcium, magnesium, ALP, glucose, amylase, lipase, Urea/BUN, CA 19-9 on treatment: worst CTC grade per patient (Table 52)
- Total bilirubin, AST, ALT, LDH, serum creatinine, chloride, sodium, albumin, potassium, calcium, magnesium, ALP, amylase, lipase during follow-up: worst CTC grade per patient (**Table 53**)

#### 7.7.2.3 Thyroid Function Tests

- TSH, T3 free, T3 total, T4 free, T4 total on treatment (Table 54)
- TSH, T3 free, T3 total, T4 free, T4 total during follow-up (Table 55)

#### 7.7.2.3 Coagulation

- PT, INR, PTT on treatment (**Table 56**)
- PT, INR, PTT during follow-up (Table 57)

#### 7.7.3 Other Safety

#### 7.7.3.1 ECG

Cardiac function of patients is evaluated as clinically indicated by ECG during protocol treatment with results reported on Treatment Report.

• Number of patients by normal or abnormal ECG, by treatment group (Table 58)

#### 7.7.3.2 Urinalysis

Dipstick urinalysis is performed as clinically indicated during protocol treatment . with results reported on Treatment Report.

• Results of urinalysis, by treatment group (Table 59)

## 7.7.4 Deaths on Study/Adverse Events Leading to Discontinuations of Protocol Treatment

- Deaths during treatment or within 4 weeks of last protocol treatment: number
  of patients who died and cause of death from Date/Cause of Death Section of
  Death Report (Table 60)
- Number of patients with adverse events leading to discontinuations of protocol treatment as identified from Off Protocol Treatment Adverse Events of End of Treatment Report (Table 61)

# 7.8 Concomitant Medications, Other Anti-Cancer Treatments, and Major Medical Problems

Investigators may prescribe concomitant medications or treatments deemed necessary to provide adequate prophylactic or supportive care. Administration of any other anticancer therapy for pancreatic cancer is not permitted while the patient is receiving protocol therapy. Thereafter, patients may be treated at the investigator's discretion. Major medical problems are those thought unrelated to protocol treatment.

- Concomitant medications during or 4 weeks after protocol treatment (reported on Treatment Report and 4-Week Post-Treatment Follow-Up Report) (**Table 62**)
- Other anti-cancer treatments for pancreatic cancer during or 4 weeks after protocol treatment (reported on Treatment Report and 4 Weeks 4-Week Post-Treatment Follow-Up Report) (**Table 63**)
- Other anti-cancer treatments for pancreatic cancer during follow-up (reported on Follow-up Report or Short Follow-up Reports) (Table 63)

• Major medical problem during or 4 weeks after protocol treatment (reported on Treatment Report and 4-Week Post-Treatment Follow-Up Report) (**Table 64**)

#### 7.9 Quality of Life

The quality of life of patients in this study is assessed at 4, 8, 12, 16 and 24 weeks from randomization during protocol treatment and then every 3 months until PD or the initiation of another chemotherapy treatment by using EORTC QLQ-C30 (version 3.0). The following are the scoring algorithms for this instrument.

#### **7.9.1 EORTC QLQ-C30**

The EORTC core questionnaire, QLQ-C30 (version 3.0), consists of five Functional Scales, Global Health Status, and nine Symptoms Scales. Each scale in the questionnaire will be scored (0 to 100) according to the EORTC recommendations in the EORTC QLQ-C30 Scoring Manual. The scoring method is summarized below. In this summary Qi refers to the ith question on the QLQ-C30.

#### Functional scale's scores:

| • Physical functioning: | (1 - ((Q1+Q2+Q3+Q4+Q5)/5 -1)/3) * 100 |
|--------------------------|---------------------------------------|
| • Role functioning: | (1 - ((Q6+Q7)/2-1)/3) * 100 |
| • Emotional functioning: | (1 - ((Q21+Q22+Q23+Q24)/4-1)/3) * 100 |
| • Cognitive functioning: | (1 - ((Q20+Q25)/2-1)/3) * 100 |
| • Social functioning: | (1 - ((Q26+Q27)/2-1)/3) * 100 |

#### Global health status score:

• Global health status/QOL: ((Q29+Q30)/2-1)/6 \* 100

#### Symptom scale's scores:

| • Fatigue: | ((Q10+Q12+Q18)/3-1)/3 * 100 |
|----------------------------------------|-----------------------------|
| <ul><li>Nausea and vomiting:</li></ul> | ((Q14+Q15)/2-1)/3 * 100 |
| • Pain: | ((Q9+Q19)/2-1)/3 * 100 |
| • Dyspnea: | ((Q8-1)/3 * 100 |
| • Insomnia: | (Q11-1)/3 * 100 |
| • Appetite loss: | (Q13-1)/3 * 100 |
| • Constipation: | (Q16-1)/3 * 100 |
| • Diarrhea: | (Q17-1)/3 * 100 |
| • Financial difficulties: | (Q28-1)/3 * 100 |

Missing items in a scale will be handled by the methods outlined in the scoring manual. In particular, values will be imputed for missing items by "assuming that the missing items have values equal to the average of those items which are present" for any scale in which at least half the items are completed. A scale in which less than half of the items are completed will be treated as missing.

#### 7.9.2 Data Sets

The analyses of quality of life data will be restricted to randomized patients who have a measurement at baseline and at least one measurement after baseline.

#### 7.9.3 Compliance

Compliance will be described, by time of evaluation, by the number and percentage of subjects who filled out a questionnaire (per subject, at least one question answered) in that period of evaluation. The denominator used in calculating the percentage for baseline will be all randomized subjects. The denominator used for all other time points will be the number of subjects known to be alive at the start of the time period (**Table 65**).

#### 7.9.4 Primary Analyses of QOL

The primary endpoints for the comparison of QOL between treatment arms will be proportions of patients who had deterioration in physical function and Global Health Status at 8 weeks and 16 weeks after the randomization. The deterioration is defined as a change score from baseline which is –10 points or lower [6]. Fisher's exact test will be used to compare the proportions of patients with deterioration between two treatment arms at these two time points (**Table 66**). No multiple adjustment for these comparisons will be made.

The proportions of patients who had improving (defined as change score from baseline of 10 points or higher) or stable (defined as change score from baseline of between – 10 and 10 points) physical function and Global Health Status at 8 weeks and 16 weeks after the randomization will also be compared between two treatment arms using Fisher's exact test **(Table 66)**.

The time to definitive deterioration in physical function and Global Health Status is defined as the time from randomization until the change score from baseline is -10 points or lower. For patients whose change scores are always higher than -10 points, the time to definitive deterioration will be censored at their last QoL assessment times. The log-rank test will be used to compare the time to definitive deterioration between two treatment arms (**Table 67**).

#### 7.9.5 Baseline and Change Score Analysis

Descriptive statistics for EORTC QOL score (mean, standard deviation) will be presented for each scale at baseline. The same statistics will be generated at each time of post-baseline evaluation. The comparability of mean baseline scores and change scores at each time of post-baseline evaluation between treatment groups will be assessed using a Wilcoxon rank sum test (**Table 68** and **Table 69**).

#### 7.9.6 **QOL Response Analysis**

QOL response for functional scales and global health status is calculated as follows: A change score of 10 points from baseline is defined as clinically relevant. Patients are considered to have clinical improvement if reporting a score 10-points or better than baseline at any time of QOL assessment. Conversely, patients are considered worsened if reporting a score minus 10-points or worse than baseline at any time of QOL assessment without any improvement. Patients whose scores are between 10-point changes from baseline at every QOL assessment will be considered as stable. In contrast to functional scales, for the determination of patient's QOL response, classification of patients into improved and worsened categories is reversed for symptom scales. A Chi-square test will then be performed to compare the distributions of these three categories between two arms (**Table 70**).

## 8. Appendices

## **Appendix 1: Tables and Figure**

**Table 1: Patient Disposition** 

| Data set: All Randomized Patients | | | |
|---|---|---|---|
| | Number of patients (%) | | |
| | G+N+D+T G+N Tota | | |
| Randomized | N=*** | N=*** | N=*** |
| Treated | *** (**) | *** (**) | *** (**) |
| On study | *** (**) | *** (**) | *** (**) |
| Off study <sup>(1)</sup> | *** (**) | *** (**) | *** (**) |
| Never Treated | *** (**) | *** (**) | *** (**) |

<sup>(1)</sup> Off all study therapies.

**Table 2: Follow-up of Patients** 

| Data set: All R | andomized Patients | | |
|--------------------------|------------------------|---------|---------|
| | Number of patients (%) | | |
| | G+N+D+T | G+N | Total |
| Number of patients alive | *** (%) | *** (%) | *** (%) |
| Follow-up (months) | | | |
| median | ** | ** | ** |
| Minimum-maximum | **_** | **_** | **_** |

**Table 3: Accrual by Center** 

Data set: All Randomized Patients Number of patients (%) G+N+D+T G+N Total N = \*\*\* N = \*\*\* \*\*\* (\*\*) \*\*\* (\*\*) \*\*\* (\*\*) Center #1 Center #2 \*\*\* (\*\*) Center #3 \*\*\* (\*\*) \*\*\* (\*\*) \*\*\* (\*\*)

Table 4: Accrual by Stratification Factor at Randomization

| Data s | set: All Randomized Patients | | |
|---|---|---|---|
| | Number | Number of patients (%) | |
| | G+N+D+T<br>N = *** | G+N<br>N=*** | Total<br>N = *** |
| Performance Status | | | |
| ECOG 0 | ** (**) | ** (**) | ** (**) |
| ECOG 1 | ** (**) | ** (**) | ** (**) |
| Prior adjuvant therapy | | | |
| Yes | ** (**) | ** (**) | ** (**) |
| No | ** (**) | ** (**) | ** (**) |

Source: Centralized Randomization File

Figure 1: Accrual by Calendar Time



Table 5: Eligibility and Reasons for Ineligibility and Major Protocol Violations

| Data se | t: All Randomized Patients | } | |
|---|---|---|---|
| | Numb | er of Patients (% | (o) |
| | G+N+D+T | G+N | Total |
| | N=*** | N=*** | N=*** |
| Eligible | *** (**) | *** (**) | *** (**) |
| Not Eligible | *** (**) | *** (**) | *** (**) |
| Reason for ineligibility | | | |
| <reason 1=""></reason> | ** | ** | ** |
| <reason 2=""></reason> | ** | ** | ** |
| | ** | ** | ** |
| Major protocol violation | | | |
| <pre><violation 1="" type=""></violation></pre> | ** | ** | ** |
| <violation 2="" type=""></violation> | ** | ** | ** |

Table 6: Treatment as Randomized Versus as Treated

| Data set: A | ll Randomized Patients | | |
|--------------------|------------------------|-----------------|----------|
| | Number | of Patients (%) | |
| | Rando | Randomized Arm | |
| | G+N+D+T | G+N | Total |
| | N=*** | N=*** | N=*** |
| Treatment received | | | |
| All G+N+D+T | *** (**) | *** (**) | *** (**) |
| Durvalumab only | *** (**) | *** (**) | *** (**) |
| Tremelimumab only | *** (**) | *** (**) | *** (**) |
| G+N Only | *** (**) | *** (**) | *** (**) |
| Not treated | *** (**) | *** (**) | *** (**) |

**Table 7: Pretreatment Characteristics at Baseline** 

| Data set: All Rand | | of patients (%) | |
|---|---|---|---|
| | G+N+D+T | G+N | Total |
| | N=*** | N=*** | N=*** |
| Gender | ( ماد ماد ) | ale ale (ale ale) | ( ماد ماد ) ماد ماد |
| Female<br>Male | ** (**)<br>** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| | ( ) | | ( ) |
| Race<br>White | ** (**) | ** (**) | ** (**) |
| Black or African American | ** (**) | ** (**) | ** (**) |
| | ** (**) | ** (**) | ** (**) |
| Age (years) | | , , | |
| N | ** | ** | ** |
| Median | ** | ** | ** |
| Min - Max | ** _ ** | ** - ** | ** _ ** |
| < 65 | ** (**) | ** (**) | ** (**) |
| ≥ 65 | ** (**) | ** (**) | ** (**) |
| ECOG Performance Status | | | |
| 0 | ** (**) | ** (**) | ** (**) |
| 1 | ** (**) | ** (**) | ** (**) |
| BSA (m <sup>2</sup> ) | | | |
| N | ** | ** | ** |
| Median | ** | ** | ** |
| Min - Max | ** _ ** | ** _ ** | ** _ ** |
| Months from initial diagnosis to randomization | | | |
| N | ** | ** | ** |
| Median | ** | ** | ** |
| Min - Max | ** _ ** | ** _ ** | ** _ ** |
| Metastatic disease at initial diagnosis | | | |
| Yes | **(**) | **(**) | ** (**) |
| No | **(**) | **(**) | **(**) |
| Months from diagnosis of metastatic disease | | | |
| following completion of prior surgical/adjuvant | | | |
| therapy | | | |
| N | ** | ** | ** |
| Median | ** | ** | ** |
| Min - Max | ** _ ** | ** - ** | ** _ ** |

**Table 8: Prior Surgery** 

| Data set | : All Randomized Patients | | |
|---|---|---|---|
| | Number | Number of Patients (%) | |
| | G+N+D+T<br>N=*** | G+N<br>N=*** | Total<br>N=*** |
| Prior surgery | | | |
| No | *** (**) | *** (**) | *** (**) |
| Yes | *** (**) | *** (**) | *** (**) |
| Procedure / Site | | | |
| Procedure / Site 1 | *** (**) | *** (**) | *** (**) |
| Procedure / Site 2 | *** (**) | *** (**) | *** (**) |
| | *** (**) | *** (**) | *** (**) |

**Table 9: Prior Radiotherapy** 

| | <del>-</del> - | | |
|---|---|---|---|
| Data set: | All Randomized Patients | | |
| | Number of patie | ents (%) | |
| | G+N+D+T<br>N=*** | G+N<br>N=*** | Total<br>N=*** |
| Any Prior Radiotherapy<br>No<br>Yes | *** (**)<br>*** (**) | *** (**)<br>*** (**) | *** (**)<br>*** (**) |
| Site of any prior radiotherapy <sup>(1)</sup><br>Site #1<br>Site #2 | *** (**)<br>*** (**)<br>*** (**) | *** (**) *** (**) ***(**) | *** (**)<br>*** (**)<br>***(**) |

<sup>(1)</sup> Patient may have more than one site of radiotherapy

**Table 10: Prior Systemic Therapy** 

| Data set: All Ra | ndomized Patients | | |
|---|---|---|---|
| | Number of | of patients (%) | |
| | G+N+D+T<br>N=*** | G+N<br>N=*** | Total<br>N=*** |
| With at least one prior systemic therapy | *** (**) | *** (**) | *** (**) |
| Type of prior systemic therapy At least one adjuvant At least one neo-adjuvant At least one metastatic | *** (**)<br>*** (**)<br>*** (**) | *** (**)<br>*** (**)<br>*** (**) | *** (**)<br>*** (**)<br>*** (**) |
| Specific drug/agent <sup>(1)</sup> | | | |
| Drug/agent #1<br>Drug/agent #2 | *** (**)<br>*** (**)<br>*** (**) | *** (**)<br>*** (**)<br>*** (**) | *** (**) *** (**) *** (**) |

<sup>(1)</sup> Patient may have more than one drug/agent.

**Table 11: Extent of Disease (Target Lesions)** 

| Data set: All Rar | ndomized Patients | | |
|---|---|---|---|
| | Number of Patients with Target Lesions (%) | | |
| | G+N+D+T | G+N | Total |
| | N=*** | N=*** | N=*** |
| Presence of Target Lesions | | | |
| Patients with at least one target lesion | *** (**) | *** (**) | *** (**) |
| Number of Target Lesions | | | |
| 1 | *** (**) | *** (**) | *** (**) |
| 2 | *** (**) | *** (**) | *** (**) |
| 3 | *** (**) | *** (**) | *** (**) |
| 4 | *** (**) | *** (**) | *** (**) |
| 5 | *** (**) | *** (**) | *** (**) |
| Largest Target Lesion in cm | | | |
| < 2 | *** (**) | *** (**) | *** (**) |
| 2-5 | *** (**) | *** (**) | *** (**) |
| > 5-10 | *** (**) | *** (**) | *** (**) |
| > 10 | *** (**) | *** (**) | *** (**) |
| Site of Target Lesion <sup>(1)</sup> | | | |
| Abdomen | *** (**) | *** (**) | *** (**) |
| Adrenals | *** (**) | *** (**) | *** (**) |
| Bone | *** (**) | *** (**) | *** (**) |
| Brain | *** (**) | *** (**) | *** (**) |
| Liver | *** (**) | *** (**) | *** (**) |
| Lung | *** (**) | *** (**) | *** (**) |
| Nodes | *** (**) | *** (**) | *** (**) |
| Pleura | *** (**) | *** (**) | *** (**) |
| Skin | *** (**) | *** (**) | *** (**) |
| Subcutaneous Tissue | *** (**) | *** (**) | *** (**) |
| | *** (**) | *** (**) | *** (**) |

<sup>(1)</sup> Patients may have target lesions at more than one site

Table 12: Extent of Disease (Non-Target Lesions)

| Data Set. A | All Randomized Patients | Number of Patients (%) | |
|---|---|---|---|
| | | 1 | 1 |
| | G+N+D+T $N=***$ | G+N | Total |
| | | N=*** | N=*** |
| Patients with no-target lesion | *** (**) | *** (**) | *** (**) |
| Site of non-target lesion <sup>(1)</sup> | | | |
| Abdomen | *** (**) | *** (**) | *** (**) |
| Adrenals | *** (**) | *** (**) | *** (** |
| Bone | *** (**) | *** (**) | *** (** |
| Brain | *** (**) | *** (**) | *** (** |
| Liver | *** (**) | *** (**) | *** (** |
| Lung | *** (**) | *** (**) | *** (** |
| Nodes | *** (**) | *** (**) | *** (** |
| Pleura | *** (**) | *** (**) | *** (** |
| Skin | *** (**) | *** (**) | *** (** |
| Subcutaneous Tissue | *** (**) | *** (**) | *** (** |
| Other | *** (**) | *** (**) | *** (**) |
| Number of non-target lesions | | | |
| 1 | *** (**) | *** (**) | *** (** |
| 2 | *** (**) | *** (**) | *** (** |
| 3 | *** (**) | *** (**) | *** (** |
| 4 | *** (**) | *** (**) | *** (** |
| ≥5 | *** (**) | *** (**) | *** (** |

<sup>(1)</sup> Patients may have non-target lesions at more than one site

**Table 13: Baseline Signs and Symptoms** 

| Data | set: All Ra | indomized F | Patients (G+) | N+D+T Arn | n) | |
|---|---|---|---|---|---|---|
| | | | | of patients (<br>N=*** | (%) | |
| | | | Worst grad | e | | Any grade |
| | NR | 1 | 2 | 3 | 4 | |
| Patients with any sign/symptom at baseline | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with particular sign or symptom, within body system: | | | | | | |
| Body System 1 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(`** |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| Body System 2 <sup>(1)</sup> | | ( ) | ( ) | · / | ( ) | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |

<sup>(1)</sup> Patients may have more than one event within a body system

## NOTE: Same table to be made for G+N Arm

**Table 14: Baseline Hematology** 

| | | Data set: All Randomized P | ationts | |
|---|---|---|---|---|
| | | | ata set: All Randomized Patients Number of Patients (%) | |
| | | G+N+D+T | G+N | Total |
| | | N = *** | N = *** | N=*** |
| Hemog | alohin | 11 | 14 - * * * | 11- |
| Ticino | Grade 0 | ** (**) | ** (**) | ** (**) |
| | Grade 1 | | | |
| | Grade 2 | ** (**)<br>** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| | | ** (**)<br>** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Platele | Not reported (1) | ** (**) | ** (**) | ** (**) |
| riateie | | ** (**) | ** (**) | ** (**) |
| | Grade 0 | ** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| | Grade 1 | ** (**) | ** (**) | ** (**) |
| HIDO | Not reported (1) | ** (**) | ** (**) | ** (**) |
| WBC | 0 10 | ** (**) | ** (**) | ** (**) |
| | Grade 0 | ** (**) | ** (**) | ** (**) |
| | Grade 1 | ** (**) | ** (**) | ** (**) |
| | Grade 2 | ** (**) | ** (**) | ** (**) |
| | Grade 3 | ** (**) | ** (**) | ** (**) |
| | Grade 4 | ** (**) | ** (**) | ** (**) |
| | Not reported (1) | ** (**) | ** (**) | ** (**) |
| Neutro | | | | |
| | Grade 0 | ** (**) | ** (**) | ** (**) |
| | Grade 1 | ** (**) | ** (**) | ** (**) |
| | Not reported (1) | ** (**) | ** (**) | ** (**) |
| Lymp | phocytes | | | |
| | Grade 0 | ** (**) | ** (**) | ** (**) |
| | Grade 1 | ** (**) | ** (**) | ** (**) |
| | Grade 2 | ** (**) | ** (**) | ** (**) |
| | Grade 3 | ** (**) | ** (**) | ** (**) |
| | Grade 4 | ** (**) | ** (**) | ** (**) |
| | Not reported (1) | ** (**) | ** (**) | ** (**) |
| RBC | 1 | | , , | , |
| | Normal | ** (**) | ** (**) | ** (**) |
| | High (2) | ** (**) | ** (**) | ** (**) |
| | Not reported (1) | ** (**) | ** (**) | ** (**) |
| Monoc | | | ( ) | ( ) |
| | Normal | ** (**) | ** (**) | ** (**) |
| | High (2) | ** (**) | ** (**) | ** (**) |
| | Not reported (1) | ** (**) | ** (**) | ** (**) |
| Eosino | | | ( ) | ( ) |
| Losine | Normal | ** (**) | ** (**) | ** (**) |
| | High <sup>(2)</sup> | ** (**) | ** (**) | ** (**) |
| | Not reported (1) | ** (**) | ** (**) | ** (**) |
| Dacon! | - | () | [ [ | () |
| Basop | Normal | ** (**) | ** (**) | ** (**) |
| | | ** (**)<br>** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| | High (2) | ** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| | Not reported (1) | ** (**) | ** (**) | ** (**) |

<sup>(1)</sup> Not done or outside the 14-day window prior to start of therapy
(2) High than upper lower limit

**Table 15: Baseline Chemistry** 

| $ \begin{array}{ c c c c } \hline & Number of Patients (\%) \\ \hline & G+N+D+T \\ N=*** & N=*** & N=*** \\ \hline \hline Total bilirubin \\ Grade 0 & **(**) & **(**) & **(**) \\ Grade 1 & **(**) & **(**) & **(**) \\ Grade 2 & **(**) & **(**) & **(**) \\ Not reported (!) & **(**) & **(**) & **(**) \\ \hline Creatinine clearance \\ Grade 0 & **(**) & **(**) & **(**) \\ Grade 1 & **(**) & **(**) & **(**) \\ Grade 1 & **(**) & **(**) & **(**) \\ Grade 2 & **(**) & **(**) & **(**) \\ Grade 3 & **(**) & **(**) & **(**) \\ Not reported (!) & **(**) & **(**) & **(**) \\ \hline ALT & Grade 0 & **(**) & **(**) & **(**) \\ Grade 1 & **(**) & **(**) & **(**) \\ Not reported (!) & **(**) & **(**) & **(**) \\ \hline AST & Grade 0 & **(**) & **(**) & **(**) \\ Grade 1 & **(**) & **(**) & **(**) \\ Not reported (!) & **(**) & **(**) & **(**) \\ Not reported (!) & **(**) & **(**) & **(**) \\ \hline LDH & Normal & **(**) & **(**) & **(**) & **(**) \\ High (!) & **(**) & **(**) & **(**) & **(**) \\ Serum Creatinine & Grade 0 & **(**) & **(**) & **(**) & **(**) \\ Grade 1 & **(**) & **(**) & **(**) & **(**) \\ Hypernatremia & Grade 0 & **(**) & **(**) & **(**) & **(**) \\ Grade 1 & **(**) & **(**) & **(**) & **(**) & **(**) \\ Grade 2 & **(**) & **(**) & **(**) & **(**) & **(**) \\ Grade 3 & **(**) & **(**) & **(**) & **(**) & **(**) \\ Hyponatremia & Grade 4 & **(**) & **(**) & **(**) & **(**) & **(**) \\ Hyponatremia & **(**) & **(**) & **(**) & **(**) & **(**) & **(**) & **(**) \\ Hyponatremia & **(**) $ | Σ |
|---|---|
| Total bilirubin Grade 0 **(**) Grade 1 **(**) Grade 2 **(**) Not reported (1) Creatinine clearance Grade 0 **(**) Grade 1 **(**) **(**) **(**) **(**) **(**) **(**) Creatinine clearance Grade 0 Grade 1 **(**) Grade 2 **(**) Grade 2 **(**) Grade 3 **(**) Not reported (1) **(**) **( | |
| Total bilirubin Grade 0 Grade 1 Grade 2 **(**) Grade 2 **(**) Not reported (1) Creatinine clearance Grade 1 **(**) Grade 2 **(**) **(**) **(**) **(**) **(**) **(**) Creatinine clearance Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) Grade 2 **(**) Grade 3 **(**) **(* | |
| Grade 0 Grade 1 Grade 2 Not reported (1) Creatinine clearance Grade 2 Grade 3 Grade 1 Grade 1 Grade 0 Grade 0 Grade 1 Grade 0 Grade 1 Grade 1 Grade 1 Grade 1 Grade 1 Grade 1 Grade 1 Grade 2 First order o | |
| Grade 1 Grade 2 Not reported (1) Creatinine clearance Grade 0 Grade 2 **(**) Grade 1 **(**) Grade 1 **(**) Grade 1 **(**) Grade 1 **(**) Grade 1 **(**) Grade 2 **(**) Grade 2 **(**) Grade 3 **(**) | otal bilirubin |
| Grade 2 Not reported (1) Creatinine clearance Grade 0 Grade 1 Grade 2 Grade 2 Grade 2 Grade 3 Grade 4 Not reported (1) ALT Grade 0 Grade 1 Grade 0 ** (**) ** (** | Grade 0 |
| Not reported (1) Creatinine clearance Grade 0 | Grade 1 |
| Creatinine clearance Grade 0 | Grade 2 |
| Grade 0 | Not reported (1) |
| Grade 1 | eatinine clearance |
| Grade 1 | Grade 0 |
| Grade 2 Grade 3 Grade 4 Not reported (1) ALT Grade 0 Grade 1 Sorte (**) Fortal (**) F | Grade 1 |
| Grade 3 Grade 4 Not reported (1) ALT Grade 0 **(**) Grade 1 **(**) **(**) Grade 1 **(**) Grade 1 **(**) Grade 0 **(**) AST Grade 0 **(**) Grade 1 **(**) Formal **(**) Not reported (1) **(**) Grade 1 **(**) **(**) **(**) **(**) **(**) **(**) **(**) Grade 1 **(**) **( | Grade 2 |
| Grade 4 Not reported (1) ALT Grade 0 ** (**) Not reported (1) AST Grade 1 ** (**) Grade 1 ** (**) AST Grade 0 ** (**) Grade 1 ** (**) AST Grade 1 ** (**) Grade 1 ** (**) ** (**) ** (**) AST Grade 1 ** (**) Grade 1 ** (**) ** (** | Grade 3 |
| Not reported (1) ALT Grade 0 Grade 1 Not reported (1) AST Grade 0 ** (**) AST Grade 0 ** (**) Grade 1 ** (**) AST Grade 0 ** (**) Grade 1 ** (**) ** (**) ** (**) ** (**) ** (**) AST Grade 1 ** (**) Not reported (1) ** (**) ** (* | Grade 4 |
| ALT Grade 0 Grade 1 Not reported (1) AST Grade 0 ** (**) Grade 1 ** (**) Grade 1 ** (**) Grade 1 ** (**) Grade 1 ** (**) ** | Not reported (1) |
| Grade 1 Not reported (1) AST Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) **(* | |
| Grade 1 Not reported (1) AST Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) **(* | Grade 0 |
| AST Grade 0 Grade 1 Not reported (1) Not reported (1) Not reported (1) Normal High(2) Not reported (1) Serum Creatinine Grade 0 ** (**) Grade 1 ** (**) Grade 1 ** (**) | |
| Grade 0 | |
| Grade 0 | |
| Grade 1 Not reported (1) Normal High(2) Not reported (1) Serum Creatinine Grade 0 Grade 1 Not reported (1) Figh (2) F | |
| Not reported (1) Normal Normal High(2) Not reported (1) Serum Creatinine Grade 0 Grade 1 Not reported (1) Hypernatremia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Not reported (1) ** (**) | |
| Normal | |
| Normal | |
| High(2) | |
| Not reported (1) | |
| Serum Creatinine Grade 0 ** (**) Grade 1 ** (**) Not reported (1) Hypernatremia Grade 0 ** (**) Grade 1 ** (**) ** (**) ** (**) ** (**) ** (**) Grade 1 ** (**) ** (**) ** (**) ** (**) ** (**) ** (**) Grade 3 Grade 4 ** (**) Not reported (1) ** (**) | _ |
| Grade 0 | - |
| Grade 1 | |
| Not reported (1) | |
| Hypernatremia Grade 0 ** (**) Grade 1 ** (**) | |
| Grade 0 | |
| Grade 1 | = |
| Grade 2 ** (**) ** (**) ** (**) Grade 3 ** (**) ** (**) ** (**) Grade 4 ** (**) ** (**) ** (**) Not reported (1) ** (**) ** (**) ** (**) | |
| Grade 3 ** (**) ** (**) ** (**) Grade 4 ** (**) ** (**) ** (**) Not reported (1) ** (**) ** (**) ** (**) | |
| Grade 4 ** (**) ** (**) ** (**) Not reported (1) ** (**) ** (**) ** (**) | |
| Not reported (1) | |
| | _ |
| Grade 2 ** (**) ** (**) ** (**) ** (**) | |
| Grade 3 ** (**) ** (**) ** (**) ** (**) | |
| Grade 4 ** (**) ** (**) ** (**) | |
| Not reported (1) | |
| Hyperkalemia | = |
| Grade 0 ** (**) ** (**) ** (**) ** (**) | |
| Grade 1 ** (**) ** (**) ** (**) | |
| Grade 2 ** (**) ** (**) ** (**) ** (**) | |
| Grade 3 ** (**) ** (**) ** (**) | |
| Grade 4 ** (**) ** (**) ** (**) | |
| Not reported (1) | |
| Hypokalemia | /рокатетта |

| Grade 0 | ** (**) | ** (**) | ** (**) |
|---|---|---|---|
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Hypercalcemia | ` / | , , | ` ' |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Hypocalcemia | | ( ) | ( ) |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| | | () | () |
| Hypermagnesemia<br>Grade 0 | ** (**) | ** (**) | ** (**) |
| | | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 1 | ** (**)<br>** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 2 | ** (**) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Hypomagnesemia | (ماد ماد ) ماد ماد | ale ale ( ale ale ) | ( ماد ماد ) . ماد ماد |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Hyperglycemia | | | |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Hypoglycemia | | | |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Hyperalbuminemia | | | ( ) |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Hypoalbuminemia | | | ( ) |
| 11ypoaiouiiiiiciiiia | I | ı l | |

| Grade 0 | ** (**) | ** (**) | ** (**) |
|---------------------|---------|---------|---------|
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Chloride | | | |
| Normal | ** (**) | ** (**) | ** (**) |
| High (2) | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Amylase | | | , |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| ALP | | , | |
| Normal | ** (**) | ** (**) | ** (**) |
| High <sup>(2)</sup> | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Lipase | | , | |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |
| Urea/BUN | | , | |
| Grade 0 | ** (**) | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) | ** (**) |

<sup>(1)</sup> Not done or outside the 14-day window prior to start of therapy
(2) High than upper lower limit

**Table 16: Baseline Thyroid Function Tests** 

| Data set: All Randomized Patients | | | |
|---|---|---|---|
| | Numl | ber of Patients (%) | |
| | G+N+D+T | G+N | Total |
| | N = *** | N = *** | N = *** |
| TSH | | | |
| Normal | ** (**) | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) | ** (**) |
| T3 Free | | | |
| Normal | ** (**) | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) | ** (**) |
| T3 Total | | | |
| Normal | ** (**) | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) | ** (**) |
| T4 Free | | | |
| Normal | ** (**) | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) | ** (**) |
| T4 Total | | | |
| Normal | ** (**) | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) | ** (**) |

**Table 17: Baseline Coagulation Tests** 

| | Data set: All Randomize | d Patients | |
|---------|-------------------------|------------|---------|
| | Number of Patients (%) | | |
| | G+N+D+T | G+N | Total |
| | N = *** | N = *** | N = *** |
| PT | | | |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| INR | , , | | ` ' |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |
| PTT | . , | | ` ' |
| Grade 1 | ** (**) | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) | ** (**) |

**Table 18: Baseline ECG** 

| Data set: All Randomized Patients | | | |
|---|---|---|---|
| | Number of patients (%) | | |
| | G+N+D+T<br>N=*** | G+N<br>N=*** | Total<br>N=*** |
| Baseline ECG: Results | | | |
| Normal | *** (**) | *** (**) | *** (**) |
| Abnormal | *** (**) | *** (**) | *** (**) |
| ECG not performed | *** (**) | *** (**) | *** (**) |

**Table 19: Baseline Urinalysis** 

| Data set: All Randomized Patients | | | |
|---|---|---|---|
| | Number of patients (%) | | |
| | G+N+D+T | G+N | Total |
| | N=*** | N=*** | N=*** |
| Urinalysis – SPOT Test | | | |
| Negative/trace | **(**) | **(**) | **(**) |
| 1+(>20 mg/dL-30 mg/dL) | **(**) | **(**) | **(**) |
| 2+(>30 mg/dL-100 mg/dL) | **(**) | **(**) | **(**) |
| 3+(>100 mg/dL-300 mg/dL) | **(**) | **(**) | **(**) |
| 4+(>300 mg/dL) | **(**) | **(**) | **(**) |
| Urinalysis – 24-Hour Test (g/day) | | | |
| Grade | | | |
| 1 | **(**) | **(**) | **(**) |
| 2 | **(**) | **(**) | **(**) |
| 3 | **(**) | **(**) | **(**) |
**Table 20: Concomitant Medications at Baseline** 

| D | ata set: All Randomized | Patients | |
|---|---|---|---|
| | Nu | Number of patients (%) | |
| | G+N+D+T N=*** | G+N<br>N=*** | Total<br>N=*** |
| Any concomitant medication (1) | | | |
| No | ** (**) | ** (**) | ** (**) |
| Yes | ** (**) | ** (**) | ** (**) |

<sup>(1)</sup>Any medication taken within 14 days prior to randomization.

Table 21: Major Medical Problems at Baseline

| Data set: All Rand | lomized Patients | | |
|---|---|---|---|
| | Number of patients (%) | | |
| | G+N+D+T | G+N | Total |
| | N = *** | N = *** | N=*** |
| Patients with at least one past or current major medical problem | ** (**) | ** (**) | ** (**) |
| Medical Problem <sup>(1)</sup> | | | |
| (from highest to lowest in frequency) | | | |
| Diabetes | ** (**) | ** (**) | ** (**) |

<sup>(1)</sup> patients may report more than one medical problem reported

**Table 22: Number of Patients by Cycle** 

| | | Number of Par | Number of Patients (%) |
|-------|-----|---------------|------------------------|
| | | G+N+D+T Arm | G+N Arm |
| Cycle | 1 | ** (**) | ** (**) |
| - | 2 | ** (**) | ** (**) |
| | 3 | ** (**) | ** (**) |
| | ••• | | |

**Table 23**: Number of Cycles of Protocol Therapy per Patient

| | Data Set: All Treated Patients | S |
|-------------------|--------------------------------|---------|
| | G+N+D+T Arm | G+N Arm |
| Number of Cycles: | | |
| N | *** | *** |
| Median | * | * |
| Min – Max | * _ * | * _ * |
| Min – Max | T = T | ጥ _ ጥ |

**Table 24: Total Treatment Duration** 

| Data Set: All Treated Patients | | | | | | |
|---|---|---|---|---|---|---|
| | | G+N+1 | D+T Arm | | G+N | Arm |
| | Durva- | Tremeli- | Gemcita- | Nab- | Gemcita- | Nab- |
| | lumab | mumab | bine | paclitaxel | bine | paclitaxel |
| Duration in weeks | | | | | | |
| N | *** | *** | *** | *** | *** | *** |
| Median | * | * | * | * | * | * |
| Min – Max | * _ * | * _ * | * _ * | * _ * | * _ * | * _ * |

Table 25: Dose Reduction, Omission or Delay and Infusion Interruption

| | Dat | ta Set: All Tre | ated Patients | | | |
|---|---|---|---|---|---|---|
| | Number of patients (%) | | | | | |
| | | G+N+ | D+T Arm | | G+N | Arm |
| | Durvalu-<br>mab<br>(N=***) | Tremeli-<br>mumab<br>(N=***) | Gemcita-<br>bine<br>(N=***) | Nab-<br>paclitaxel<br>(N=***) | Gemcita-<br>bine<br>(N=***) | Nab-<br>paclitaxel<br>(N=***) |
| At least one dose reduction Reason for dose reduction: | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <reason 1=""></reason> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <reason 2=""></reason> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| At least one dose omission Reason for dose omission: | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <pre><reason 1=""></reason></pre> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <reason 2=""></reason> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| At least one dose delay<br>Reason for delay: | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <reason 1=""></reason> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <reason 2=""></reason> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| At least one infusion interruption Reason for interruption: | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <reason 1=""></reason> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| <reason 2=""></reason> | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |

**Table 26: Cumulative Dose** 

| | | Data Set: | All Treated P | atients | | |
|---|---|---|---|---|---|---|
| | | G+N+1 | D+T Arm | | G+N | Arm |
| | Durva- | Tremeli- | Gemcita- | Nab- | | |
| | lumab | mumab | bine | paclitaxel | bine | paclitaxel |
| Cumulative dose<br>N | *** | *** | *** | *** | *** | *** |
| Mean (STD)<br>Median | ** (**)<br>* | ** (**)<br>* | ** (**)<br>* | ** (**)<br>* | ** (**)<br>* | ** (**)<br>* |
| Min – Max | * _ * | * _ * | * _ * | * _ * | * _ * | * _ * |

**Table 27: Dose Intensity** 

| Data Set: All Treated Patients | | | | | | |
|---|---|---|---|---|---|---|
| | | G+N+1 | D+T Arm | | G+N | G+N Arm |
| | Durva- | Tremeli- | Gemcita- | Nab- | | |
| | lumab | mumab | bine | paclitaxel | bine | paclitaxel |
| Dose Intensity N Mean (STD) Median Min – Max | *** ** (**) * * _ * | *** ** (**) * * - * | ***<br>** (**)<br>*<br>* _ * | *** ** (**) * * - * | *** ** (**) * * _ * | *** ** (**) * *_* |

**Table 28: Relative Dose Intensity** 

| | Data Set: All Treated Patients | | | | | |
|---|---|---|---|---|---|---|
| | | G+N+D | +T Arm | | G+N | G+N Arm |
| | Durvalumab<br>(N=***) | Tremelimumab (N=***) | Gemcitabine (N=***) | Nab-<br>paclitaxel<br>(N=***) | Gemcitabine (N=***) | Nab-<br>paclitaxel<br>(N=***) |
| Relative Dose intensity | | | | | | |
| ≥ 90% planned intensity | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| $\geq 80\%$ - $< 90\%$ planned intensity | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| $\geq 60\% - < 80\%$ planned intensity | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| < 60% planned intensity | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |

**Table 29: Off Treatment Summary** 

| | | Data Se | t: All Treated Pat | ients | | |
|---|---|---|---|---|---|---|
| | | G+N+D+T | Arm | | G+N | G+N Arm |
| | Durvalumab<br>(N=***) | Tremelimumab<br>(N=***) | Gemcitabine (N=***) | Nab-<br>paclitaxel<br>(N=***) | Gemcitabine (N=***) | Nab-<br>paclitaxel<br>(N=***) |
| Off treatment | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Reason off treatment | | | | | | |
| Treatment Completed | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Progressive disease (objective) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Symptomatic progression | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Intercurrent Illness –<br>adverse events<br>unrelated to protocol<br>treatment | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Adverse events related to protocol therapy | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patient Refusal (not related to adverse | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| event)<br>Death | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Other reason | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |

**Table 30: All Deaths** 

| Data set: All Randomized Patients | | |
|---|---|---|
| | Number of Pa | atients (%) |
| | G+N+D+T | G+N |
| | N=*** | N=*** |
| Number of Patients who died | ** (**) | ** (**) |
| Cause of Death | | |
| Pancreatic cancer only | ** | ** |
| Toxicity from protocol treatment | ** | ** |
| Pancreatic cancer + Toxicity from protocol treatment complication | ** | ** |
| Non-protocol Treatment Complication | ** | ** |
| Colorectal cancer + Non-protocol Treatment Complication | ** | ** |
| Other Primary Malignancy | ** | ** |
| Other Condition or Circumstance | ** | ** |

Figure 2: Kaplan-Meier Curves for Overall Survival



Table 31: Log Rank and Cox Regression Model for Overall Survival

| | Da | ta set: All F | Randomized Pation | ents | • | • |
|---|---|---|---|---|---|---|
| | N | Uni | Multivariate Analysis <sup>(2)</sup> | | | |
| Treatment Arm/ | | Median | Hazard | Log- | Hazard | P-value |
| Prognostic Factors at | | Survival | Ratio <sup>(4)</sup> | rank | Ratio <sup>(4)</sup> | from Cox |
| Baseline | | (Months) | (90% CI) | p-value | (90% C.I.) | model |
| Treatment arm | | | | 0.*** | | 0.*** |
| G+N+D+T | *** | ** ** | **.** | | **.** | |
| G+N | *** | **.** | (**.**,**.**) | | (**.**,**.**) | |
| Gender | | | | 0.*** | | 0.*** |
| Male | *** | **.** | NC (3) | | **.** | |
| Female | *** | **.** | | | (**.**,**.**) | |
| Age | | | | 0.*** | | 0.*** |
| <65 | *** | **.** | NC | | **.** | |
| ≥65 | *** | **.** | | | (**.**,**.**) | |
| Number of organ sites | | | | 0.*** | | 0.*** |
| ≤ 2 | *** | **.** | NC | | **.** | |
| >2 | *** | ** ** | | | (**.**,**.**) | |

<sup>(1)</sup> Stratified; (2) Stratified Cox regression with all factors included; (3) NC = not computed (4) Hazard ratio of first category over second category

**Table 32: Survival by Subsets** 

| | Da | ata set: | All Randomized P | atients | | |
|---|---|---|---|---|---|---|
| | | | G+N+D+T | | G+N | |
| | | | Median | | Median | Hazard Ratio <sup>(1)</sup> |
| Factors | Value | N | Survival | N | Survival | 90% C.I. |
| | | | (90% C.I.) | | (90% C.I.) | |
| Performance Status | ECOG 0 | ** | **.** | ** | **.** | ** ** |
| at baseline | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | ECOG 1 | ** | **.** | ** | **.** | ** ** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Age | <65 | ** | **.** | ** | **.** | **.** |
| S | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | ≥65 | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Gender | Female | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | Male | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Race | White | ** | ** ** | ** | **.** | ** ** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | Black | ** | ** ** | ** | **.** | ** ** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | Other | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Number of organ | ≤2 | ** | **.** | ** | **.** | **.** |
| sites | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | >2 | ** | ** ** | ** | ** ** | ** ** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |

<sup>(1)</sup> G+N+D+T over G+N hazard ratio (Unstratified)

**Table 33: Progression Summary** 

| | Number of l | Patients (%) |
|----------------------------------------|------------------|--------------|
| | G+N+D+T<br>N=*** | G+N<br>N=*** |
| Patients who progressed | *** (**) | *** (**) |
| Progression on protocol treatment | ** | ** |
| Progression off protocol treatment | ** | ** |
| Death (without documented progression) | ** | ** |
| Patients who were censored | *** (**) | *** (**) |
| Reason Censored | | |
| Lost to follow-up | ** | ** |
| Not progressed | ** | ** |

Figure 3: Kaplan-Meier Curves for Progression Free Survival



Table 34: Log Rank and Cox Regression Model for Progression Free Survival (PFS)

| | Da | ata set: All F | Randomized Pation | ents | | |
|---|---|---|---|---|---|---|
| | N | Univariate Analysis <sup>(1)</sup> | | | Multivariate Analysis <sup>(2)</sup> | |
| Treatment Arm/ | | Median | Hazard | Log- | Hazard | P-value |
| Prognostic Factors at | | PFS | Ratio <sup>(4)</sup> | rank | Ratio <sup>(4)</sup> | from Cox |
| Baseline | | (Months) | (90% CI) | p-value | (90% C.I.) | model |
| Treatment arm | | | | 0.*** | | 0.*** |
| G+N+D+T | *** | ** ** | **.** | | **.** | |
| G+N | *** | ** ** | (**.**,**.**) | | (**.**,**.**) | |
| Gender | | | | 0.*** | | 0.*** |
| Male | *** | **.** | NC (3) | | ** ** | |
| Female | *** | **.** | | | (**.**,**.**) | |
| Age | | | | 0.*** | | 0.*** |
| <65 | *** | **.** | NC | | ** ** | |
| ≥65 | *** | **.** | | | (**.**,**.**) | |
| Number of organ sites | | | | 0.*** | | 0.*** |
| <i>≤</i> 2 | *** | **.** | NC | | ** ** | |
| >2 | *** | **.** | | | (**.**,**.**) | |

<sup>(1)</sup> Stratified; (2) Stratified Cox regression with all factors included; (3) NC = not computed

Note: Same table will be made for sensitivity analyses which (1) censor the patients who have received other anti-cancer treatments prior to documentation of disease relapse/progression or death at the earliest time when these treatments began or (2) treat them as having PFS events at the earliest time when these treatments began.

<sup>(4)</sup> Hazard ratio of first category over second category

Table 35: Progression Free Survival (PFS) by Subsets

| | Da | ata set: | All Randomized P | atients | | |
|---|---|---|---|---|---|---|
| | | | G+N+D+T | | G+N | |
| | | | Median | | Median | Hazard Ratio <sup>(1)</sup> |
| Factors | Value | N | Survival | N | Survival | 90% C.I. |
| | | | (90% C.I.) | | (90% C.I.) | |
| Performance Status | ECOG 0 | ** | **.** | ** | **.** | ** ** |
| at baseline | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | ECOG 1 | ** | ** ** | ** | ** ** | ** ** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Age | <65 | ** | ** ** | ** | ** ** | ** ** |
| <i>8</i> - | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | ≥65 | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Gender | Female | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | Male | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Race | White | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | Black | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | Other | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| Number of organ | ≤2 | ** | ** ** | ** | ** ** | ** ** |
| sites | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |
| | >2 | ** | **.** | ** | **.** | **.** |
| | | | (**.**,**.**) | | (**.**,**.**) | (**.**,**.**) |

<sup>(1)</sup> G+N+D+T over G+N hazard ratio (Unstratified)

**Table 36: Treatment Objective Response** 

Data set: All Randomized Patients

| Data set: A | Data set: All Randomized Patients | |
|---|---|---|
| | Number of Pat | ients (%) <sup>a</sup> |
| | N=*** | |
| | G+N+D+T N=*** | G+N |
| | | N=*** |
| Patients with at least one target lesion | N=*** | N=*** |
| Response-evaluable | N=*** | N=*** |
| Complete response (CR) | ** (**) | ** (**) |
| Partial response (PR) | ** (**) | ** (**) |
| Stable disease (SD) | ** (**) | ** (**) |
| Progressive disease (PD) | ** (**) | ** (**) |
| Inevaluable for response (IN) | ** (**) | ** (**) |
| <reason 1=""></reason> | ** | ** |
| <reason 2=""></reason> | ** | ** |
| Not response evaluable | N=*** | N=*** |
| Never treated | ** | ** |
| Not assessed (NA) | ** | ** |
| Patients with no target lesions | N=*** | N=*** |
| Progressive disease (PD) | ** | ** |
| Inevaluable for response (IN) | ** | ** |
| <reason 1=""></reason> | ** | ** |
| <reason 2=""></reason> | ** | ** |
| Not assessed (NA) | ** | ** |
| Never treated | ** | ** |

<sup>&</sup>lt;sup>a</sup> percentages are calculated out of the number of randomized patients

Table 37: Cochran Mantel Haenszel and Logistic Regression Model for Objective Response

| | | Data set: All Rando | omized Patients | S | |
|---|---|---|---|---|---|
| | | Univariate A | analysis <sup>(1)</sup> | Multivariat | e Analysis (2) |
| Treatmen | nt/ Prognostic Factors | Odds Ratio <sup>(4)</sup><br>(90%CI) | CMH<br>p-value | Odds Ratio <sup>(4)</sup><br>(90% C.I.) | p-value<br>from logistic<br>regression |
| Treatment a $G^+$ | orm<br>-N+D+T: G+N | ** **<br>(** .**,**.**) | 0.*** | **.**<br>(**.**,**.**) | 0.*** |
| Gender Ma | ale: Female | NC (3) | 0.*** | **.**<br>(**.**,**.**) | 0.*** |
| Age <6 | 75: ≥65 | NC | 0.*** | **.**<br>(**.**,**.**) | 0.*** |
| Number of o ≤2. | organ sites : >2 | NC | 0.*** | **.**<br>(**.**,**.**) | 0.*** |

<sup>(1)</sup> Stratified
(2) Stratified Logistic regression, all factors included
(3) NC = not computed
(4) Odds ratio of first category over second category

**Table 38: Objective Response According to Pretreatment Characteristics** 

| Da | ta set: All Randomized Patients | |
|---|---|---|
| | Number of Objective Respon | nses/Number of Patients (%) |
| | G+N+D+T | G+N |
| | N=*** | N=*** |
| Gender | | |
| Male | **/** (**) | **/** (**) |
| Female | **/** (**) | **/** (**) |
| Age | | |
| < 65 years | **/** (**) | **/** (**) |
| ≥65 years | **/** (**) | **/** (**) |
| Race | | |
| White | **/** (**) | **/** (**) |
| Black | **/** (**) | **/** (**) |
| Other | **/** (**) | **/** (**) |
| Baseline performance status | ` ' | |
| ECOG 0-1 | **/** (**) | **/** (**) |
| ECOG 2 | **/** (**) | **/** (**) |
| Number of organ sites | ` ' | |
| ≤2 | **/** (**) | **/** (**) |
| >2 | **/** (**) | **/** (**) |

**Table 39: Duration of Objective Response** 

| Data set: All Random | nized Patients with CR of | or PR | |
|---|---|---|---|
| | G+N+D+T | G+N | P-value <sup>(1)</sup> |
| | N=*** | N=*** | |
| Median Duration of Objective Response (months) | *** | *** | .** |
| (90% CI) | (**-**) | (**-**) | |

<sup>(1)</sup> Stratified

**Table 40: Immune Response (iRECIST)** 

Data set: All Randomized Patients Number of Patients (%)<sup>a</sup> N=\*\*\* G+N+D+T G+N N=\*\*\* N=\*\*\* Patients with at least one target lesion N=\*\*\* N=\*\*\* Response-evaluable N=\*\*\* N=\*\*\* Immune Complete response (iCR) \*\* (\*\*) \*\* (\*\*) Immune Partial response (iPR) \*\* (\*\*) \*\* (\*\*) Immune Stable disease (iSD) \*\* (\*\*) \*\* (\*\*) \*\* (\*\*) Immune confirmed progression (iCPD) Immune unconfirmed progression (iUPD) Inevaluable for response (IN) <Reason 1> <Reason 2> N=\*\*\* N=\*\*\* Not response evaluable \*\* \*\* Never treated \*\* Not assessed (NA) Patients without any target lesion N=\*\*\* N=\*\*\* Immune confirmed progression (iCPD) Immune unconfirmed progression (iUPD) Inevaluable for response (IN) <Reason 1> \*\* \*\* <Reason 2> Not assessed (NA) Never treated

<sup>&</sup>lt;sup>a</sup> percentages are calculated out of the number of randomized patients

Table 41: Cochran Mantel Haenszel and Logistic Regression Model for Immune Response

| | | Data set: All Rando | omized Patients | S | |
|---|---|---|---|---|---|
| | | Univariate A | nalysis <sup>(1)</sup> | Multivariate | e Analysis (2) |
| Treatment/ I | Prognostic Factors | Odds Ratio <sup>(4)</sup><br>(90%CI) | CMH<br>p-value | Odds Ratio <sup>(4)</sup><br>(90% C.I.) | p-value<br>from logistic<br>regression |
| Treatment arm $G+N-$ | +D+T: G+N | ** **<br>(** .**, ** .**) | 0.*** | ** **<br>(** .** ,** .**) | 0.*** |
| Gender <i>Male:</i> | Female | NC <sup>(3)</sup> | 0.*** | **.**<br>(**.**,**.**) | 0.*** |
| Age <65: | ≥65 | NC | 0.*** | ** .**<br>(** .** ,** .**) | 0.*** |
| Number of org ≤2: > | | NC | 0.*** | **.**<br>(**.**,**.**) | 0.*** |

<sup>(1)</sup> Stratified
(2) Stratified Logistic regression, all factors included
(3) NC = not computed
(4) Odds ratio of first category over second category

**Table 42: Immune Response According to Pretreatment Characteristics** 

| Da | ata set: All Randomized Patients | |
|---|---|---|
| | Number of Immune Respons | ses/Number of Patients (%) |
| | G+N+D+T | G+N |
| | N=*** | N=*** |
| Gender | | |
| Male | **/** (**) | **/** (**) |
| Female | **/** (**) | **/** (**) |
| Age | , , | . , |
| < 65 years | **/** (**) | **/** (**) |
| ≥65 years | **/** (**) | **/** (**) |
| Race | | |
| White | **/** (**) | **/** (**) |
| Black | **/** (**) | **/** (**) |
| Other | **/** (**) | **/** (**) |
| Baseline performance status | , , | . , |
| ECOG 0-1 | **/** (**) | **/** (**) |
| ECOG 2 | **/** (**) | **/** (**) |
| Number of organ sites | | |
| ≤ 2 | **/** (**) | **/** (**) |
| >2 | **/** (**) | **/** (**) |

**Table 43: Duration of Immune Response** 

| Data set: All Rando | mized Patients with iCR or | · iPR | |
|---|---|---|---|
| | G+N+D+T | G+N | P-value <sup>(1)</sup> |
| | N=*** | N=*** | |
| Median Duration of Immune Response (months) | *** | *** | .** |
| (90% CI) | (**-**) | (**-**) | |

<sup>(1)</sup> Stratified

**Table 44: Acute (On Treatment) Adverse Events** 

| | | | | of patients ( | %) | | |
|---|---|---|---|---|---|---|---|
| | | | | N=*** | | | |
| | | | Worst g | grade | | | Any<br>grade |
| | NR | 1 | 2 | 3 | 4 | 5 | |
| Patients with any AE | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE within | | | | | | | |
| category | | | | | | | |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 1 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) | **(** |

<sup>(1)</sup> Patients may have more than one event within a category.

Note: Same table will be made for patients on G+N Arm.

**Table 45: Severe Acute (On Treatment) Adverse Events** 

| Data set: All Tre | ated Patients on C | G+N+D+T | Arm | |
|---|---|---|---|---|
| | Number of patients (%) N=*** | | | |
| | Worst | Any grade 3 or higher AE | | |
| | 3 | 4 | 5 | |
| Patients with any AE | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE within category | | | | |
| Category 1 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) |

<sup>(1)</sup> Patients may have more than one event within a category.

Note: Same table will be made for patients on G+N Arm.

**Table 46: Drug Related Acute (on Treatment) Adverse Events** 

# (1) Related to Durvalumab

| Da | ta set: All Tre | eated Patients | on G+N+D+ | T Arm | | |
|---|---|---|---|---|---|---|
| | | N | Number of pa<br>N=** | tients (%) | | |
| | | W | orst grade | | | Any grade |
| | 1 | 2 | 3 | 4 | 5 | |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE related to durvalumab within category | | | | | | |
| Category 1 <sup>(a)</sup> | | | | | | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| ••• | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(a)</sup> | | | | | | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |

<sup>(</sup>a) Patients may have more than one event within a category.

# (2) Related to Tremelimumab

| Data | set: All Tre | ated Patients | on G+N+D+ | T Arm | | |
|---|---|---|---|---|---|---|
| | | | Number of p<br>N=* | | | |
| | | | Any grade | | | |
| | 1 | 2 | 3 | 4 | 5 | |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE related to | | | | | | |
| Tremelimumab within category | | | | | | |
| Category 1 <sup>(a)</sup> | | | | | | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(a)</sup> | . , | ` / | , , | ` / | ` / | . , |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |

<sup>(</sup>a) Patients may have more than one event within a category.

## (3) Related to Durvalumab or Tremelimumab

| Data | set: All Tre | ated Patients | on G+N+D+ | T Arm | | |
|---|---|---|---|---|---|---|
| | | | Number of p<br>N=* | | | |
| | | | Any grade | | | |
| | 1 | 2 | 3 | 4 | 5 | |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE related to<br>Durvalumab or Tremelimumab<br>within category | | | | | | |
| Category 1 <sup>(a)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(a)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |

<sup>(</sup>a) Patients may have more than one event within a category.

## (4) Related to Both Durvalumab and Tremelimumab

| Data | set: All Tre | ated Patients | on G+N+D+ | T Arm | | |
|---|---|---|---|---|---|---|
| | Number of patients (%) N=*** | | | | | |
| | | V | Vorst grade | | | Any grade |
| | 1 | 2 | 3 | 4 | 5 | |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE related to both<br>Durvalumab and<br>Tremelimumab within category | | | | | | |
| Category 1 <sup>(a)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(a)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |

### (5) Related to Gemcitabine

| Dat | ta set: All Tre | eated Patients | on G+N+D+ | T Arm | | |
|---|---|---|---|---|---|---|
| | | N | Number of pa<br>N=** | | | |
| | | W | orst grade | | | Any grade |
| | 1 | 2 | 3 | 4 | 5 | |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE related to | | | | | | |
| Gemecitabine within category | | | | | | |
| Category 1 <sup>(a)</sup> | | | | | | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(a)</sup> | , , | , | , | , | , , | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |

<sup>(</sup>a) Patients may have more than one event within a category.

Note: Same table will be made for patients on G+N Arm.

(6) Related to Nab-paclitaxel

| Data | set: All Tre | ated Patients | on G+N+D+ | T Arm | | |
|---|---|---|---|---|---|---|
| | Number of patients (%) N=*** | | | | | |
| | | V | Vorst grade | | | Any grade |
| | 1 | 2 | 3 | 4 | 5 | |
| | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with AE related to | | | | | | |
| Nab-paclitaxel within category | | | | | | |
| Category 1 <sup>(a)</sup> | | | | | | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(a)</sup> | | | • | , í | | |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| ••• | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |

<sup>(</sup>a) Patients may have more than one event within a category.

Note: Same table will be made for patients on G+N Arm.

Table 47: Immune-related Acute (On Treatment) Adverse Events

| | Data set: | All Treated | Patients on | G+N+D+T | Arm | |
|---|---|---|---|---|---|---|
| | | Number of patients (%) N=*** | | | | |
| | | | Worst grade | | | Any grade |
| | 1 | 2 | 3 | 4 | 5 | |
| Patients with any irAE | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with irAE | | | | | | |
| within category | | | | | | |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 1 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| ••• | | , | , | . , | , , | , |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | | | | | · | |

<sup>(1)</sup> Patients may have more than one event within a category.

Note: Same table will be made for patients on G+N Arm.

**Table 48: Severe Acute (On Treatment) Immune-related Adverse Events** 

| | Number of patients (%)<br>N=*** | | | |
|---|---|---|---|---|
| | Wors | t grade | | Any grade 3 of higher irrAE |
| | 3 | 4 | 5 | |
| Patients with any irAE | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with irAE within | | | | |
| category | | | | |
| | **(**) | **(**) | **(**) | **(**) |
| Category 1 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) |

<sup>(1)</sup> Patients may have more than one event within a category.

Note: Same table will be made for patients on G+N Arm.

Table 49: Delayed (During Follow-up) Adverse Events

| | Data set: | All Treated | Patients on | G+N+D+T | Arm | |
|---|---|---|---|---|---|---|
| | | Number of patients (%) N=*** | | | | |
| | | | Worst grade | | | Any grade |
| | 1 | 2 | 3 | 4 | 5 | |
| Patients with any delayed AE | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) | ** (**) |
| Patients with delayed | | | | | | |
| AE within category | | | | | | |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 1 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 2 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 3 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Category 2 <sup>(1)</sup> | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |
| Event 1 | **(**) | **(**) | **(**) | **(**) | **(**) | **(**) |

<sup>(1)</sup> Patients may have more than one event within a category.

Note: The same type of table will be made for G+N Arm.

**Table 50: Hematology During Protocol Treatment: Worst Grade per Patient** 

| | Data set: All Treated Patients | |
|---------------------|--------------------------------|--------------|
| | Number of I | Patients (%) |
| | G+N+D+T | G+N |
| | N = *** | N = *** |
| Hemoglobin | | |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Platelet | | |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| WBC | , , , | ` / |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Neutrophils | , , , | ` ^ |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| RBC | , , , | |
| Normal | ** (**) | ** (**) |
| High <sup>(1)</sup> | ** (**) | ** (**) |
| Lymphocytes | , , , | |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Monocytes | | |
| Normal | ** (**) | ** (**) |
| High <sup>(1)</sup> | ** (**) | ** (**) |
| Eosinophils | | |
| Normal | ** (**) | ** (**) |
| High <sup>(1)</sup> | ** (**) | ** (**) |
| Basophils | | |
| Normal | ** (**) | ** (**) |
| High <sup>(1)</sup> | ** (**) | ** (**) |

<sup>(1)</sup> Greater than upper normal limit

**Table 51: Hematology During Follow-up: Worst Grade per Patient** 

| Data set: All Treated Patients | |
|---|---|
| | of Patients (%) |
| G+N+D+T | G+N |
| N = *** | N = *** |
| ** (**) | ** (**) |
| ** (**) | ** (**) |
| | ** (**) |
| ** (**) | ** (**) |
| , , , | . , |
| ** (**) | ** (**) |
| ** (**) | ** (**) |
| | ** (**) |
| | ** (**) |
| ** (**) | ** (**) |
| | ** (**) |
| | ** (**) |
| | ** (**) |
| ** (**) | ** (**) |
| ` / | ** (**) |
| ` ' | ** (**) |
| ` / | ** (**) |
| ** (**) | ** (**) |
| | ** (**) |
| ** (**) | ** (**) |
| | ** (**) |
| | ** (**) |
| ` / | ** (**) |
| ** (**) | ** (**) |
| ` / | ** (**) |
| | ( ) |
| ** (**) | ** (**) |
| | ** (**) |
| | ( ) |
| ** (**) | ** (**) |
| | ** (**) |
| | Number G+N+D+T N = *** ** (**) ** (**) ** (**) ** (**) |

<sup>(1)</sup> Greater than upper normal limit

Table 52: Serum Chemistry during Protocol Treatment: Worst Grade per Patient

| Data set: All Treated Patients | | |
|--------------------------------|------------------------|--------------------|
| | Number of Patients (%) | |
| | <u> </u> | |
| | G+N+D+T<br>N = *** | G+N<br>N = *** |
| Total bilirubin | 11 - | 14 - |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Creatinine clearance | | ( ) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | |
| Grade 4 | ** (**) | ** (**)<br>** (**) |
| Not reported (1) | ** (**) | ** (**)<br>** (**) |
| ALT | (11) | (**) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Not reported (1) | ` / | |
| AST | ** (**) | ** (**) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | | |
| | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Not reported (1)<br>LDH | ** (**) | ** (**) |
| Normal | ** (**) | ** (**) |
| High <sup>(2)</sup> | ` * | |
| Not reported (1) | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Serum Creatinine | (11) | (**) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hypernatremia | (11) | (**) |
| Grade 0 | ** (**) | ** (**) |
| Grade 0<br>Grade 1 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 1 Grade 2 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 3 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 4 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hyponatremia Crode 0 | ** (**) | ** (**) |
| Grade 0 | ** (**) | ** (**)<br>** (**) |
| Grade 1 | ** (**) | ** (**)<br>** (**) |
| Grade 2 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 3 | ** (**) | ** (**)<br>** (**) |
| Grade 4 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hyperkalemia | ** (**/ | ** (**) |
| Grade 0 | ** (**) | ** (**)<br>** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |

| 1 (1) | 1 | |
|--------------------|--------------------|---------------------|
| Not reported (1) | ** (**) | ** (**) |
| Hypokalemia | 4.5.74.5 | t.t. 71.15 |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hypercalcemia | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hypocalcemia | 4.5.74.5 | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hypermagnesemia | distriction | dede (dede) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hypomagnesemia | ** (**) | ske ske ( ske ske ) |
| Grade 1 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 1<br>Grade 2 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 3 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Grade 4 | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hyperglycemia | | ( ) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hypoglycemia | ( ) | ( ) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hyperalbuminemia | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| | • • | |

| NI ( 1(1) | 44 (44) | |
|------------------|---------|------------|
| Not reported (1) | ** (**) | ** (**) |
| Hypoalbuminemia | ** (**) | ** (**) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Chloride | A. (A.) | h.t. (1.1) |
| Normal | ** (**) | ** (**) |
| High (2) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Amylase | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| ALP | | |
| Normal | ** (**) | ** (**) |
| High (2) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Lipase | , , | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Urea/BUN | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |

<sup>(1)</sup> Greater than upper normal limit

Table 53: Serum Chemistry During Follow-up: Worst Grade per Patient

| I | Data set: All Treated Patients | D (* (0/) |
|---------------------------|--------------------------------|---------------|
| | Number of I | Patients (%) |
| | G+N+D+T G+N | |
| | N = *** | N = *** |
| Total bilirubin | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Creatinine clearance | · / | ` / |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| ALT | ( ) | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| AST | ( ) | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Not reported (1) | | ** (**) |
| | ** (**) | () |
| LDH Normal | ** (**) | ** (**) |
| Normal | ** (**) | ** (**) |
| High <sup>(2)</sup> | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Serum Creatinine | deale (deale) | abada (abada) |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hypernatremia | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hyponatremia | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Hyperkalemia <sup>1</sup> | . / | , , |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |

| Grade 0 | II la la maia | 1 | |
|---|---|---|---|
| Grade 1 | Hypokalemia | ** (**) | ** (**) |
| Grade 2 Grade 3 Grade 4 Five series of the s | | ` ' | |
| Grade 3 | | 1 1 | |
| Grade 4 | | | |
| Not reported (1) Hypercalcemia Grade 0 Grade 1 Grade 2 **(**) Grade 2 **(**) Grade 3 **(**) Frade 3 Grade 0 **(**) Hypocalcemia Grade 0 **(**) **(**) **(**) **(**) **(**) Hypocalcemia Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) Grade 2 **(**) Grade 2 **(**) Grade 3 **(**) Grade 3 **(**) Grade 1 **(**) **(**) Hypermagnesemia Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) Grade 2 **(**) Grade 3 **(**) Grade 1 **(**) Grade 3 **(**) Grade 4 **(**) Not reported (1) **(**) Hypomagnesemia Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) **(**) Hypomagnesemia Grade 0 **(**) Grade 1 **(**) Grade 3 **(**) Grade 4 **(**) Not reported (1) **(**) Hyperglycemia Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) Grade 2 **(**) Grade 1 **(**) **(**) Hyperglycemia Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) **(**) Hypoplycemia Grade 0 **(**) Grade 1 **(**) Grade 1 **(**) **(**) Hypoplycemia Grade 0 **(**) Hypoglycemia Grade 1 **(**) Grade 1 **(**) Grade 1 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 1 **(**) Grade 1 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 1 **(**) Grade 1 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 1 **(**) Grade 1 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 1 **(**) Grade 1 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 1 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 0 **(**) Hypoglycemia Grade 1 **(**) Hypoglycemia Grade 1 **(**) Hypoglycemia Grade 2 **(**) Hypoglycemia Grade 3 **(**) Hypoglycemia Grade 4 **(**) Hypoglycemia Grade 1 **(**) Hypoglycemia Grade 1 **(**) Hypoglycemia Grade 1 **(**) Hyp | | | |
| Hypercalcemia Grade 0 | | | |
| Grade 0 | | ** (**) | ** (**) |
| Grade 1 Grade 2 Grade 3 Grade 4 Reference 2 Grade 3 Grade 4 Reference 3 Grade 4 Reference 3 Grade 6 Grade 1 Reference 3 Grade 2 Reference 3 Reference | | district (district | aleade (aleade) |
| Grade 2 Grade 3 Grade 4 Set (**) Grade 4 Not reported (1) Hypocalcemia Grade 1 Grade 2 Grade 2 Grade 1 Grade 2 Grade 2 Grade 3 Grade 4 Set (**) Grade 2 Grade 3 Grade 4 Set (**) Grade 3 Grade 4 Set (**) Grade 3 Grade 4 Set (**) Hypermagnesemia Grade 0 Grade 1 Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Hypermagnesemia Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Grade 2 Grade 3 Grade 4 Set (**) Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Hypomagnesemia Grade 4 Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Hypomagnesemia Grade 0 Grade 1 Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Grade 1 Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Hyporeptod (1) Hyperglycemia Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Hyperglycemia Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Hyporglycemia Grade 2 Grade 3 Grade 4 Set (**) Grade 1 Grade 2 Grade 3 Grade 4 Set (**) Hyporglycemia Grade 2 Grade 3 Grade 4 Set (**) Hyporglycemia Grade 4 Set (**) Grade 5 Grade 6 Grade 1 Grade 1 Grade 2 Set (**) Hyporglycemia Grade 4 Set (**) Hyporglycemia Grade 4 Set (**) Hyporglycemia Grade 4 Set (**) Hyporglycemia Grade 6 Grade 1 Set (**) Hyporglycemia Grade 1 Set (**) Hyporglycemia Grade 2 Set (**) Hyporglycemia Grade 3 Set (**) Hyporglycemia Grade 4 Set (**) Hyporglycemia Grade 4 Set (**) Hyporglycemia Grade 6 Grade 1 Set (**) Hyporglycemia Grade 1 Set (**) Hyporglycemia Grade 2 Set (**) Hyporglycemia Grade 3 Set (**) Hyporglycemia Grade 4 Set (**) Hyporglycemia Grade 4 Set (**) Hyporglycemia Grade 6 Set (**) Hyporglycemia Grade 7 Set (**) Hyporglycemia Grade 9 Set (**) Hyporglycemia Grade 1 Set (**) Hyporglycemia Grade 1 Set (**) Hyporglycemia | | 3 7 | |
| Grade 3 Grade 4 Not reported (1) Hypocalcemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hyporoalcemia Grade 1 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hypermagnesemia Grade 0 Grade 1 Standard 1 Grade 0 Grade 1 Grade 0 Grade 1 Warehald 1 | | | |
| Grade 4 ** (**) ** (**) ** (**) Hypocalcemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) Hypermagnesemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Hypermagnesemia Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Hypomagnesemia Grade 4 ** (**) ** (**) Grade 1 ** (**) ** (**) Hypomagnesemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Hypomagnesemia Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Hyporglycemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) | | | |
| Not reported (1) Hypocalcemia Grade 0 Grade 0 Grade 1 Grade 2 Grade 2 Grade 3 Grade 4 Not reported (1) Hypermagnesemia Grade 2 Grade 1 Grade 0 Grade 0 Grade 0 Grade 0 Grade 1 Grade 0 Grade 1 Grade 2 Fixe in the state of the state of the state of the state of the state of Grade of the | | | |
| Hypocalcemia Grade 0 | | 1 | |
| Grade 0 Grade 1 Grade 2 Grade 2 Grade 2 Grade 3 Grade 4 Not reported (1) Hypomagnesemia Grade 4 Grade 1 Grade 1 Grade 2 Grade 3 Grade 4 First Sorred 4 First Sorred 5 Grade 1 Grade 1 Grade 2 First Sorred 5 Grade 3 First Sorred 5 Grade 4 First Sorred 6 First Sorred 6 First Sorred 7 Grade 1 First Sorred 7 Grade 1 First Sorred 8 First Sorred 8 First Sorred 9 First Sor | | ** (**) | ** (**) |
| Grade 1 Grade 2 Grade 3 Grade 3 Grade 4 Not reported (1) Hypermagnesemia Grade 4 Not reported (1) Grade 2 Grade 3 Grade 0 Grade 1 Grade 2 First (1) Grade 2 First (1) Grade 3 Grade 4 First (1) Grade 3 First (1) Grade 3 First (1) Grade 3 First (1) Grade 4 First (1) Fi | | | |
| Grade 2 Grade 3 Grade 4 Not reported (1) Hypermagnesemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 1 Grade 2 Grade 3 Grade 1 Grade 2 Grade 3 Grade 3 Grade 1 Grade 1 Grade 3 Grade 4 Figure 1 Grade 3 Grade 4 Figure 1 Grade 3 Grade 4 Figure 1 Grade 1 Grade 1 Figure 1 Grade 1 Figure 1 Grade 1 Figure 1 Grade 2 Figure 1 Grade 2 Figure 1 Grade 3 Figure 1 Grade 1 Figure 1 | | | |
| Grade 3 Grade 4 Not reported (1) Hypermagnesemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Figure 1 Grade 3 Grade 1 Grade 2 Grade 3 Grade 4 Figure 1 Grade 0 Figure 1 Grade 0 Figure 1 Grade 0 Figure 1 Grade 1 Figure 1 Grade 1 Figure 1 Grade 0 Figure 1 Figure | | | ** (**) |
| Grade 4 Not reported (1) Hypermagnesemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hypomagnesemia Grade 4 Not reported (1) Hypomagnesemia Grade 5 Grade 6 Grade 1 Grade 7 Not reported (1) Hypomagnesemia Grade 0 Grade 1 Grade 2 First (1) Grade 2 First (1) Grade 3 First (1) Grade 1 First (1) Grade 3 First (1) Grade 3 First (1) Grade 4 First (1) Grade 3 First (1) Grade 4 First (1) Grade 6 First (1) Grade 7 First (1) Grade 8 First (1) Grade 9 First (1) Grade 1 First (1) First | | | |
| Not reported (1) | | | ** (**) |
| Hypermagnesemia Grade 0 | | | ** (**) |
| Grade 0 | Not reported (1) | ** (**) | ** (**) |
| Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hypomagnesemia Grade 2 Grade 3 Grade 1 Grade 0 Grade 1 Grade 2 Grade 0 Grade 1 Grade 1 Grade 2 Fixed 3 Grade 4 Fixed 4 Fixed 5 Fixed 6 Fixed 6 Fixed 6 Fixed 7 Fixed 7 Fixed 8 Fixed 8 Fixed 8 Fixed 8 Fixed 8 Fixed 9 Fixed | Hypermagnesemia | | |
| Grade 2 Grade 3 Grade 4 Not reported (1) Hypomagnesemia Grade 1 Grade 2 Grade 2 Grade 0 Grade 1 Grade 2 Grade 3 F* (**) Grade 1 Grade 2 F* (**) Grade 3 F* (**) Grade 3 F* (**) Grade 3 F* (**) Grade 4 F* (**) F* (** | Grade 0 | ** (**) | ** (**) |
| Grade 3 Grade 4 Not reported (1) Hypomagnesemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hypomagnesemia Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hyperglycemia Grade 1 Grade 2 Grade 3 Grade 1 Grade 2 Grade 3 Grade 1 Grade 1 Grade 2 Grade 3 Grade 1 Grade 1 Grade 2 Grade 3 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hyperglycemia Grade 2 Grade 3 Grade 4 Not reported (1) Hypoglycemia Grade 4 First (**) Grade 5 Grade 6 First (**) Grade 7 Grade 8 First (**) Grade 9 First (**) Hypoglycemia Grade 0 First (**) Grade 1 First (**) | Grade 1 | ** (**) | ** (**) |
| Grade 4 Not reported (1) Hypomagnesemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hyperglycemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Figure 1 Grade 6 Grade 1 Figure 1 Grade 7 Grade 8 Grade 8 Grade 9 Grade 1 Figure 1 Grade 1 Figure 1 Grade 2 Figure 1 Grade 3 Figure 1 Grade 3 Figure 1 Grade 3 Figure 1 Grade 4 Figure 1 Figure | | ** (**) | ** (**) |
| Not reported (1) Hypomagnesemia Grade 0 Grade 1 Grade 2 ** (**) Grade 3 Grade 4 Not reported (1) Hyperglycemia Grade 2 ** (**) Grade 3 ** (**) ** (**) Hyperglycemia Grade 0 ** (**) Grade 1 ** (**) Grade 2 ** (**) Grade 3 ** (**) ** (**) ** (**) ** (**) Hypoglycemia Grade 0 ** (**) Grade 1 ** (**) Grade 3 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) Grade 1 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) Grade 1 ** (**) ** (**) Hypoglycemia Grade 1 ** (**) Grade 2 ** (**) Grade 3 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) Grade 1 ** (**) Hypoglycemia Grade 0 ** (**) | Grade 3 | ** (**) | ** (**) |
| Hypomagnesemia Grade 0 Grade 1 Grade 2 ** (**) Grade 3 ** (**) Grade 4 ** (**) Hyperglycemia Grade 0 ** (**) Grade 1 ** (**) Grade 1 ** (**) Grade 2 ** (**) Grade 1 ** (**) Grade 2 ** (**) Grade 3 ** (**) Grade 3 ** (**) Grade 4 ** (**) Hypoglycemia Grade 0 ** (**) Grade 1 ** (**) Grade 3 ** (**) ** (**) Hypoglycemia Grade 0 ** (**) Grade 1 ** (**) Grade 1 ** (**) ** (**) Hypoglycemia Grade 2 ** (**) Grade 3 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 3 ** (**) ** (**) ** (**) Hyperalbuminemia Grade 0 ** (**) Grade 1 ** (**) Grade 2 ** (**) Grade 2 ** (**) Grade 3 Grade 4 ** (**) Grade 3 Grade 4 ** (**) Grade 3 Grade 4 ** (**) Grade 3 Grade 4 ** (**) Grade 3 Grade 4 ** (**) Grade 3 ** (**) Grade 3 ** (**) ** (**) ** (**) ** (**) ** (**) Grade 3 ** (**) | | ** (**) | ** (**) |
| Grade 0 | Not reported (1) | ** (**) | ** (**) |
| Grade 1 | Hypomagnesemia | | |
| Grade 2 | Grade 0 | ** (**) | ** (**) |
| Grade 3 | Grade 1 | ** (**) | ** (**) |
| Grade 4 Not reported (1) Hyperglycemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hypoglycemia Grade 4 ** (**) Grade 3 ** (**) | Grade 2 | ** (**) | ** (**) |
| Not reported (1) | Grade 3 | ** (**) | ** (**) |
| Hyperglycemia Grade 0 | Grade 4 | ** (**) | ** (**) |
| Grade 0 | Not reported (1) | ** (**) | ** (**) |
| Grade 1 | Hyperglycemia | | |
| Grade 2 | Grade 0 | ** (**) | ** (**) |
| Grade 3 | Grade 1 | ** (**) | ** (**) |
| Grade 4 Not reported (1) Hypoglycemia Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Not reported (1) Hypoglycemia Grade 3 Grade 4 Not reported (1) Hyperalbuminemia Grade 1 Grade 2 ** (**) Hyperalbuminemia Grade 1 Grade 2 ** (**) Grade 3 ** (**) Hyperalbuminemia Grade 0 ** (**) Grade 1 Grade 2 ** (**) Grade 3 ** (**) Grade 4 ** (**) Grade 5 Grade 6 ** (**) Grade 7 Grade 8 ** (**) Grade 9 ** (**) ** (**) ** (**) ** (**) ** (**) | Grade 2 | ** (**) | ** (**) |
| Not reported (1) | Grade 3 | ** (**) | ** (**) |
| Hypoglycemia Grade 0 Grade 1 We will be seemed as a | | ** (**) | ** (**) |
| Grade 0 | Not reported (1) | ** (**) | ** (**) |
| Grade 1 | Hypoglycemia | | |
| Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) Not reported (1) ** (**) ** (**) Hyperalbuminemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) | Grade 0 | ** (**) | ** (**) |
| Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) Not reported (1) ** (**) ** (**) Hyperalbuminemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) | Grade 1 | ** (**) | ** (**) |
| Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) Not reported (1) ** (**) Hyperalbuminemia Grade 0 ** (**) ** (**) Grade 1 ** (**) Grade 2 ** (**) Grade 3 ** (**) Grade 4 ** (**) ** (**) | Grade 2 | ** (**) | ** (**) |
| Grade 4 ** (**) ** (**) ** (**) Hyperalbuminemia Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) Grade 3 ** (**) Grade 4 ** (**) ** (**) | Grade 3 | | |
| Not reported (1) | Grade 4 | | |
| Hyperalbuminemia ** (**) ** (**) Grade 0 ** (**) ** (**) Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) | Not reported (1) | | |
| Grade 0 | | | |
| Grade 1 ** (**) ** (**) Grade 2 ** (**) ** (**) Grade 3 ** (**) Grade 4 ** (**) ** (**) | | ** (**) | ** (**) |
| Grade 2 ** (**) ** (**) Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) | Grade 1 | | |
| Grade 3 ** (**) ** (**) Grade 4 ** (**) ** (**) | Grade 2 | | |
| Grade 4 ** (**) ** (**) | Grade 3 | | |
| | Not reported (1) | ** (**) | |

| Hypoalbuminemia | | |
|------------------|---------|---------|
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Chloride | , | |
| Normal | ** (**) | ** (**) |
| High (2) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Amylase | , , | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| ALP | | , , |
| Normal | ** (**) | ** (**) |
| High (2) | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Lipase | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |
| Urea/BUN | | |
| Grade 0 | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| Not reported (1) | ** (**) | ** (**) |

<sup>(1)</sup> Greater than upper normal limit

 Table 54: Thyroid Function Tests: Worst During Protocol Treatment

| Data | set: All Treated Patients | |
|--------------|---------------------------|------------------------|
| | Number of P | Number of Patients (%) |
| | G+N+D+T | G+N |
| | N = *** | N = *** |
| TSH | | |
| Normal | ** (**) | |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | , , | ** (**) |
| T3 Free | ** (**) | ` ' |
| Normal | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |
| T3 Total | , | ** (**) |
| Normal | ** (**) | ( ) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |
| T4 Free | , | ** (**) |
| Normal | ** (**) | ( ) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |
| T4 Total | , | ** (**) |
| Normal | ** (**) | ( ) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |

Table 55: Thyroid Function Tests: Worst during Follow-up

| | Data set: All Treated Patients | D : (0/) |
|--------------|--------------------------------|----------|
| | Number of Patients (%) | |
| | G+N+D+T | G+N |
| | N = *** | N = *** |
| TSH | | |
| Normal | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |
| T3 Free | , , | , , |
| Normal | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |
| T3 Total | , , | , |
| Normal | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |
| T4 Free | , | , |
| Normal | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |
| T4 Total | ` ´ | ` ' |
| Normal | ** (**) | ** (**) |
| <1-0.5xLLN | ** (**) | ** (**) |
| <0.5-0.1xLLN | ** (**) | ** (**) |
| <0.1xLLN | ** (**) | ** (**) |

**Table 56: Coagulation Tests: Worst During Protocol Treatment** 

| Γ | Data set: All Treated Patients | |
|---------|--------------------------------|------------------------|
| | Number of P | Number of Patients (%) |
| | G+N+D+T | G+N |
| | N = *** | N = *** |
| PT | | |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| INR | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | . , | |
| PTT | ** (**) | ** (**) |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |

**Table 57: Coagulation Tests: Worst During Follow-up** 

| | Data set: All Treated Patients | |
|---------|--------------------------------|---------|
| | Number of Patients (%) | |
| | G+N+D+T | G+N |
| | N = *** | N = *** |
| PT | | |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| INR | , , | |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |
| PTT | ` ' | |
| Grade 1 | ** (**) | ** (**) |
| Grade 2 | ** (**) | ** (**) |
| Grade 3 | ** (**) | ** (**) |
| Grade 4 | ** (**) | ** (**) |

**Table 58: ECG Results During Protocol Treatment** 

| Data set: All Treated Patients | | |
|---|---|---|
| | Number of pati | ents (%) |
| | G+N+D+T | G+N |
| | N=*** | N=*** |
| ECG reported | *** (**) | *** (**) |
| All Normal | ** | ** |
| At least one abnormal but none clinically important At least one abnormal and clinically important | ** | ** |
| ECG not reported/not performed | *** (**) | *** (**) |

**Table 59: Urinalysis During Protocol Treatment** 

| Data set: All Treated Patients | | |
|-----------------------------------|------------------------|----------|
| | Number of patients (%) | |
| | G+N+D+T | G+N |
| | N=*** | N=*** |
| Urinalysis – SPOT Test | | |
| Negative/trace | **(**) | **(**) |
| 1+(>20 mg/dL-30 mg/dL) | **(**) | **(**) |
| 2+(>30 mg/dL-100 mg/dL) | **(**) | **(`**´) |
| 3+(>100 mg/dL-300 mg/dL) | **(**) | **(**) |
| 4+(>300 mg/dL) | **(**) | **(**) |
| Urinalysis – 24-Hour Test (g/day) | | |
| Grade | | |
| 1 | **(**) | **(**) |
| 2 | **(**) | **(**) |
| 3 | **(**) | **(**) |

**Table 60: Deaths During or within 4 weeks of Last Protocol Treatment** 

| Data set: All Trea | ited Patients | |
|---|---|---|
| | Number of Patients (%) | |
| | G+N+D+T<br>N=*** | G+N<br>N=*** |
| Number of Patients who died during or within 4 weeks of last protocol treatment | ** (**) | ** (**) |
| Cause of Death | | |
| Colorectal cancer | ** | ** |
| Toxicity from protocol treatment | ** | ** |
| Colorectal cancer + Toxicity from protocol | ** | ** |
| treatment complication | | |
| Non-protocol Treatment Complication | ** | ** |
| Colorectal cancer + Non-protocol | ** | ** |
| Treatment Complication | | |
| Other Primary Malignancy | ** | ** |
| Other Condition or Circumstance | ** | ** |

Table 61: Adverse Event leading to Discontinuation of protocol Treatment<sup>(a)</sup>

| | Number of patients (%) | |
|---|---|---|
| | G+N+D+T<br>N=*** | G+N<br>N=*** |
| Number discontinued durvalumab from adverse events | ** (**) | ** (**) |
| <adverse 1="" event=""></adverse> | | |
| <adverse 2="" event=""></adverse> | ** | ** |
| | ** | ** |
| Number discontinued Tremelimunab from adverse events | ** (**) | ** (**) |
| <adverse 1="" event=""></adverse> | | |
| <adverse 2="" event=""></adverse> | ** | ** |
| | ** | ** |
| Number discontinued Gemcitabine from adverse events | *************************************** | ***(**)*) |
| <adverse 1="" event=""></adverse> | | |
| <adverse 2="" event=""></adverse> | *oklok | *** |
| | slokok: | *** |
| Number discontinued Nan-paclitaxel from adverse events | ************************************** | ***(**)*) |
| <adverse 1="" event=""></adverse> | ** | ** |
| <adverse 2="" event=""></adverse> | Holok | *** |
| | ** | ** |

<sup>(</sup>a) From End of Treatment Form with off reasons= ="Adverse events related to protocol therapy".

**Table 62: Concomitant Medications** 

| Data set: All Treated Patients | | |
|---|---|---|
| | Number of patients (%) | |
| | G+N+D+T | G+N |
| | N = *** | N=*** |
| Any concomitant medication during or 4 weeks after protocol treatment No Yes | | |
| | ** (**)<br>** (**) | ** (**)<br>** (**) |
| Type of concomitant medications <sup>(1)</sup> Medication A | ** (**) | ** (**) |

<sup>(1):</sup> patients may have received more than one concomitant medication.

**Table 63: Anti-Cancer Treatment** 

| | Number of patients (%) | |
|---|---|---|
| | G+N+D+T<br>N=*** | G+N<br>N =*** |
| Number of patients with any anti-cancer treatment during or 4 weeks after protocol treatment | *** (**) | NAP (NAP) |
| Chemotherapy <sup>(1)</sup> Drug 1 Radiotherapy <sup>(1)</sup> Hormonal therapy <sup>(1)</sup> Drug 1 | *** (**) *** (**) *** (**) *** (**) | NAP (NAP)<br>NAP (NAP)<br>NAP (NAP)<br>NAP (NAP)<br>NAP (NAP) |
| Immunotherapy <sup>(1)</sup> Drug 1 Other <sup>(1)</sup> Drug 1 | *** (**) *** (**) *** (**) *** (**) | NAP (NAP)<br>NAP (NAP)<br>NAP (NAP)<br>NAP (NAP) |
| Number of patients with any anti-cancer treatment during follow-up | *** (**) | *** (**) |
| Chemotherapy (1) Drug 1 Radiotherapy (1) Hormonal therapy (1) Drug 1 Immunotherapy (1) Drug 1 Other (1) Drug 1 | *** (**) *** (**) *** (**) *** (**) *** (**) *** (**) *** (**) | *** (**) |

<sup>(1)</sup> Patients could have more than one type of anti-cancer treatment. NA=Not applicable.

**Table 64: Major Medical Problems** 

| | Number of patients (%) | |
|---|---|---|
| | G+N+D+T G- | |
| | N = *** | N=*** |
| Any major medical problem during or 4 weeks after protocol treatment | | |
| No | | |
| Yes | | |
| | ** (**) | ** (**) |
| | ** (**) | ** (**) |
| Type of major medical problems <sup>(1)</sup> | | |
| Medication A | ** (**) | ** (**) |

<sup>(1):</sup> patients may have more than one major medical problem.

Table 65: Compliance Rate with QoL Assessment by Treatment Arm

| | G+1 | N+D+T | ( | G+N |
|---|---|---|---|---|
| | Expected | Received (%) | Expected | Received (%) |
| Baseline | *** | ** (**) | *** | ** (**) |
| During protocol treatment | | | | |
| 4 weeks | *** | ** (**) | *** | ** (**) |
| 8 weeks | *** | ** (**) | *** | ** (**) |
| 12 weeks | *** | ** (**) | *** | ** (**) |
| 16 weeks | *** | ** (**) | *** | ** (**) |
| 24 weeks | *** | ** (**) | *** | ** (**) |
| After protocol treatment | | | | , , |
| 3 months | *** | ** (**) | *** | ** (**) |
| 6 months | *** | ** (**) | *** | ** (**) |
| 12 months | *** | ** (**) | *** | ** (**) |
| 15 months | *** | ** (**) | *** | ** (**) |
| 18 months | *** | ** (**) | *** | ** (**) |
| 21 months | *** | ** (**) | *** | ** (**) |
| 24 months | *** | ** (**) | *** | ** (**) |

Table 66: Proportion of Patients with Deterioration, Improvement or Stable QoL

| | 1 | | 1 | |
|----------------------|-----|-------------|-------------|----------|
| | N | G+N+D+T | G+N | P value* |
| | 11 | N (%) | N (%) | 1 value |
| Deterioration | | | | |
| Physical function | | | | 0.*** |
| Week 8 | *** | *** (**.**) | *** (**.**) | |
| Week 16 | *** | *** (**.**) | *** (**.**) | |
| Global health status | | ` , | , , | 0.*** |
| Week 8 | *** | *** (**.**) | *** (**.**) | |
| Week 16 | *** | *** (**.**) | *** (**.**) | |
| Improvement | | | | |
| Physical function | | | | 0.*** |
| Week 8 | *** | *** (**.**) | *** (**.**) | 0. |
| Week 16 | *** | *** (**.**) | *** (**.**) | |
| Global health status | | ( . ) | ( . ) | 0.*** |
| Week 8 | *** | *** (**.**) | *** (**.**) | 0. |
| Week 16 | *** | *** (**.**) | *** (**.**) | |
| Stable | | | | |
| Physical function | | | | 0.*** |
| Week 8 | *** | *** (**.**) | *** (**.**) | 0. |
| Week 16 | *** | *** (** **) | *** (**.**) | |
| Global health status | | ( · ) | ( , ) | 0.*** |
| Week 8 | *** | *** (**.**) | *** (**.**) | 0. |
| Week 16 | *** | *** (**.**) | *** (**.**) | |

<sup>\*</sup> Fisher's exact test

**Table 67: Time to Deterioration in QoL Primary Endpoints** 

| Data set: All patients who had baseline and at least one follow-up QoL assessment | | | | |
|---|---|---|---|---|
| | ( | G+N+D+T | | G+N |
| | N | N Median (months) (90% CI) | | Median (months)<br>(90% CI) |
| Physical function | *** | **.**<br>(**.**, **.**) | *** | ** **<br>(** **, ** **) |
| Global Health Scale | *** | ** **<br>(** ** , ** .**) | *** | ** **<br>(** ** , ** .**) |

**Table 68: QoL: Summary Baseline Scores** 

| | G+N+D+T | G+N | P value* |
|----------------------|---------|-----|----------|
| Functional scales | | | |
| Physical | | | 0.*** |
| N | *** | *** | |
| Mean | *** | *** | |
| STD | *** | *** | |
| Global health status | | | 0.*** |
| N | *** | *** | |
| Mean | *** | *** | |
| STD | *** | *** | |
| Symptom scales | | | |
| Fatigue | | | 0.*** |
| N | *** | *** | |
| Mean | *** | *** | |
| STD | *** | *** | |
| | ••• | | |

<sup>\*</sup> Wilcoxon rank sum test

Table 69: Summary QOL Change Scores from Baseline for Scale/Domain/Item at Each Time Period\*

| | 0.37.5.7 | 6.33 | D. I. J. data |
|---------------------------|----------|---------|---------------|
| | G+N+D+T | G+N | P Value** |
| Scale/Domain/Item | | | |
| During protocol treatment | | | .** |
| Week 4 | | | |
| N | *** | *** | |
| Mean (STD) | ** (**) | ** (**) | |
| Week 8 | | | .** |
| N | | | |
| Mean (STD) | ** (**) | ** (**) | |
| Week 12 | | | .** |
| N | | | |
| Mean (STD) | ** (**) | ** (**) | |
| Week 16 | | | .** |
| N | | | |
| Mean (STD) | ** (**) | ** (**) | |
| Week 24 | | | .** |
| N | | | |
| Mean (STD) | ** (**) | ** (**) | |
| After protocol treatment | | | .** |
| 3 months | | | |
| N<br>M (GTD) | *** | *** | |
| Mean (STD) | ** (**) | ** (**) | ata da |
| 6 months | | | .** |
| N<br>M (GTD) | ** (**) | ** (**) | |
| Mean (STD) | ** (**) | ** (**) | ** |
| 9 months | | | .** |
| N<br>Magn (STD) | ** (**) | ** (**) | |
| Mean (STD) | ** (**) | ** (**) | ** |
| 12 months | | | |
| N<br>Magn (STD) | ** (**) | ** (**) | |
| Mean (STD) | () | () | ** |
| 15 months<br>N | | | .*** |
| | ** (**) | ** (**) | |
| Mean (STD) 18 months | (**) | ( ) | ** |
| N | | | |
| Mean (STD) | ** (**) | ** (**) | |
| 21 months | | | ** |
| N N | | | |
| Mean (STD) | ** (**) | ** (**) | |
| 24 months | | | ** |
| N N | | | |
| Mean (STD) | ** (**) | ** (**) | |
| Tricuit (DTD) | | | |

<sup>\*</sup> Table will be provided for each scale/domain/item.

\*\* Wilcoxon rank sum test

**Table 70: Results for QOL Response Analyses** 

| | | G+N+D+ | Γ | | G+N | | |
|---|---|---|---|---|---|---|---|
| Domain | Improved | Stable | Worsened | Improve | d Stable | Worsened | P-value* |
| | | N (%) | | | N (%) | | |
| EORTC QLQ-C | C30 | | | | | | |
| Physical | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Role | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Emotional | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Cognitive | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Social | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Global | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Pain | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Fatigue | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Nausea | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Dyspnea | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Sleep | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Appetite | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Constipation | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Diarrhea | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |
| Financial | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | ***(**) | .** |

<sup>\*</sup> Chi-square test